Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06

Version: 1.0, 09/MAY/2018

Page: 

Sponsor Name and Smith & Nephew Orthopaedics AG

Address: Oberneuhofstrasse 10d

6340 Baar Switzerland

Investigational SUTUREFIX ULTRA Suture Anchor

SUTUREFIX CURVED Suture Anchor

Protocol Author(s): Fiona Schlomowitsch; Mehluli Ndlovu

| Suturefix Ultra Suture Anchor Suturefix Curved Suture Anchor | > smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market 1 year Clinical | Number: 17-5010-06 |
| Follow-up Study to evaluate safety and performance of | Version: 1.0, 09/MAY/2018 |
| the SUTUREFIX ULTRA and SUTUREFIX CURVED | Page: |
| Suture Anchors in shoulder and hip arthroscopic repair | |

## 1. SIGNATURES

### 1.1 Principal Investigator Signature Page

This page will be returned to Smith & Nephew Orthopaedics AG and a copy retained at the investigational site.

I have read the attached protocol entitled I have read the attached protocol entitled", version 1.0, dated 09/MAY/2018, and agree to abide by all provisions set forth herein.

I agree to comply with the Investigator's Obligations stipulated in Section 21.4 of the protocol,
I agree to ensure that the confidential information contained in this document will not be used for
any purpose other than the conduct of the described clinical investigation without the prior
written consent of Smith & Nephew Orthopaedics AG

| Name | Signature | Date Signed<br>(DD/MMM/YYYY) |
|------|-----------|------------------------------|

| Suturefix Ultra Suture Anchor Suturefix Curved Suture Anchor | *smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market 1 year Clinical | <b>Number:</b> 17-5010-06 |
| Follow-up Study to evaluate safety and performance of | <b>Version:</b> 1.0, 09/MAY/2018 |
| the SUTUREFIX ULTRA and SUTUREFIX CURVED | Page: |
| Suture Anchors in shoulder and hip arthroscopic repair | |

# 1.2 SPONSOR APPROVAL

| Role | Approver Name | Approver Signature | Date Approved (DD/MMM/YYYY) |
|---|---|---|---|
| Head of Global Clinical | Andy Weymann for<br>Robert Eichelkraut | | |
| Operations | Robert Elcheikraut | A begun | 10/MAY/2018 |
| Head of Global Clinical | Andy Weymann for Beate Hanson | ' ' ' | |
| Strategy | Deale Hanson | A begun | 10/MAY/2018 |
| Head of Global | Alan Passington | 0 | |
| Biostatistics | Alan Rossington | Milosingho | 11/MAY/2018 |
| Head of Global Data | Alan Rossington | . 0 | |
| Sciences | Alan Rossington | Alloringh | 11/MAY/2018 |

| Suturefix Ultra Suture Anchor Suturefix Curved Suture Anchor | *smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market 1 year Clinical | Number: 17-5010-06 |
| Follow-up Study to evaluate safety and performance of | <b>Version:</b> 1.0, 09/MAY/2018 |
| the SUTUREFIX ULTRA and SUTUREFIX CURVED | Page: |
| Suture Anchors in shoulder and hip arthroscopic repair | |

# 2. SYNOPSIS

| Title of Study: | Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREELY ULTRA and SUTUREELY CURVE |
|---|---|
| | safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED |
| | Suture Anchors in shoulder and hip arthroscopic repair |
| Study Design: | Prospective |
| | Approximately 8 sites: |
| | - 4 sites for hip group |
| | - 4 sites for shoulder group |
| | Two-arms (hip and shoulder) |
| Study Type: | Post-market study |
| Study | SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchor |
| Product: | SO FORCE IN SETT CANA SO FORCE IN SOURCE SUIGNOTION |
| Study | Prospective, multicenter, post-market clinical follow-up to support CE Mark |
| Purpose: | certification and Notified Body (BSI) for the Shoulder and Hip repair indications. |
| | Data to confirm safety and performance levels acceptable for the risk benefit |
| | profile of the devices. |
| Primary | To demonstrate the performance of the SUTUREFIX ULTRA and SUTUREFIX |
| Objective: | CURVED Suture Anchors in hip and shoulder for arthroscopic treatment over a time period of 6 months after arthroscopy. |
| Secondary | To assess safety and performance, supporting the use of SUTUREFIX ULTRA |
| Objective: | and SUTUREFIX CURVED Suture Anchors in hip and shoulder arthroscopy repair. |
| Statistical | The study sample was decided based on the feasibility of recruitment, enrolment |
| Rationale: | and follow-up considerations. The study is therefore not powered for any |
| | statistical testing but will be able to estimate a success rate of 86% with a 95% |
| | confidence interval (CI) [75: 97]. Previous studies suggest that the success rate |
| | among patients who have undergone any Suture Anchors for arthroscopic |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06 Version: 1.0, 09/MAY/2018

Page: 

| | instability repair is 71-97%. |
|---|---|
| Sample Size: | A total of 80 subjects; 40 subjects for the shoulder group and 40 subjects for the hip group, will receive at least one device, SUTUREFIX ULTRA and/or SUTUREFIX CURVED Suture Anchor. A sample size of 40 subjects will estimate a success rate of 89% with a 95% confidence interval (CI) [78: 100] with 55% probability. |
| Number of<br>Study Sites: | Approximately 8 sites: • 4 sites for study hip group • 4 sites for study shoulder group |
| Targeted<br>Global<br>Regions: | Europe |

| Suturefix Ultra Suture Anchor Suturefix Curved Suture Anchor | > smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market 1 year Clinical | Number: 17-5010-06 |
| Follow-up Study to evaluate safety and performance of | Version: 1.0, 09/MAY/2018 |
| the SUTUREFIX ULTRA and SUTUREFIX CURVED | Page: |
| Suture Anchors in shoulder and hip arthroscopic repair | |

| Inclusion | All subjects |
|---|---|
| Criteria: | <ol> <li>Subject has consented to participate in the study by signing the EC-approved informed consent form</li> <li>Subject is ≥ 18 years of age at time of surgery</li> <li>Subject condition meets proposed indication to SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchor</li> <li>Subject requiring shoulder or hip arthroscopic labral repair surgery from physical findings, subject symptoms and radiographic finding</li> <li>Bone quality and quantity must be adequate to allow proper placement of the suture anchor</li> <li>Able to follow instructions.</li> <li>Willing and able to make all required study visits.</li> <li>Hip subjects</li> <li>FAI (Femoroacetabular Impingement)</li> </ol> |
| | Shoulder subjects |
| | 9. Subject with a history of recurrent dislocation/subluxation of the shoulder Hip |
| Exclusion | All subjects |
| Criteria: | <ol> <li>All subjects</li> <li>Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1 (pre-operative)</li> <li>Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures</li> <li>Any subject that meets the definition of a Vulnerable Subject per ISO14155:2011: individual whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate</li> <li>Subjects with a history of poor compliance with medical treatment</li> <li>Contraindications or hypersensitivity to the use of the SUTUREFIX ULTRA and/or SUTUREFIX CURVED Suture Anchor, or their components (e.g. silicone, polyester). Where material sensitivity is suspected, appropriate tests should be performed and sensitivity ruled out prior to implantation</li> <li>Prior ipsilateral surgeries performed on the joint space</li> <li>Pathological conditions of bone, such as cystic changes or severe osteopenia, which would compromise secure anchor fixation</li> <li>Pathological conditions in the soft tissues to be attached that would impair</li> </ol> |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Number:** 17-5010-06


Page: 

### secure fixation by suture

- 9. Comminuted bone surface, which would compromise secure anchor fixation
- 10. Physical conditions which would eliminate, or tend to eliminate, adequate anchor support or impair healing
- 11. Epileptic history

## **Hip subjects**

12. Dysplasia latera/central less than 20°

## **Shoulder subjects**

- 13. Glenoid and/or humeral bone loss considered excessive by the treating orthopaedic surgeon
- 14. MDI: Multi-directional instability
- 15. Psychosomatic voluntary shoulder subluxation

| Suturefix Ultra Suture Anchor Suturefix Curved Suture Anchor | > smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market 1 year Clinical | Number: 17-5010-06 |
| Follow-up Study to evaluate safety and performance of | Version: 1.0, 09/MAY/2018 |
| the SUTUREFIX ULTRA and SUTUREFIX CURVED | Page: |
| Suture Anchors in shoulder and hip arthroscopic repair | |

| Study | Study duration: 24 months |
|---|---|
| Duration: | Full analysis: after 12 month follow-up |
| | Enrollment period: 12 months |
| Primary endpoint: | Clinical success rate, defined as subjects without signs of failure and/or re-intervention at 6 months, as assessed by the surgeon |
| Secondary endpoint(s): | <ul> <li>Clinical success rate, defined as subjects without signs of failure and/or reintervention at 12 months, as assessed by the surgeon</li> <li>Intra-operative anchor deployment success rate</li> <li>Number of anchors pulled out</li> </ul> |
| | <ul> <li>Use of additional anchors as a result of intra operative failure</li> <li>Device-related re-intervention</li> <li>Safety evaluation at all time points</li> <li>Post-operative clinical success rate and performance assessed with subject reported outcomes as follows: <ul> <li>All subjects</li> </ul> </li> </ul> |
| | <ul> <li>Subject pain assessed with a VAS at 6 months* and 12 months*</li> <li>Subject satisfaction assessed with a VAS at 6 months* and 12 months*</li> <li>EQ-5D Questionnaire at 6 months* and 12 months*</li> </ul> |
| | Hip subjects |
| | <ul> <li>Hip Outcome Score Activities of Daily Living (HOOS-ADL) at 6 months* and 12 months*</li> <li>Modified Harris Hip Score (HHS) at 6 months* and 12 months*</li> </ul> |
| | Shoulder subjects |
| | <ul> <li>ROWE Shoulder Scores at 6 months* and 12 months*</li> <li>ASES Shoulder Scores at 6 months* and 12 months*</li> <li>Constant-Murley Shoulder Score at 6 months* and 12 months*</li> </ul> |
| | * Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference |
| Safety Data | AEs, SAEs, ADEs, SADE, USADEs |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Number:** 17-5010-06

Page: 

## **STUDY SCHEMATIC** (should be identical to Table 9.1.1-1)

| | Visit 1 | Visit 2 | Visit 3<br>Visit | Visit 4 Telephone Call or Visit | Visit 5<br>Unscheduled<br>Visit |
|---|---|---|---|---|---|
| Schedule of events (*as needed) | Pre-<br>Operative | Operative<br>through<br>Discharge | 6 Months<br>(± 1 M) | 12 Months<br>(± 1 M) | |
| Informed Consent | <b>√</b> | | | | |
| Inclusion/Exclusion Criteria | V | | | | |
| Demographics/ Medical History | <b>√</b> | | | | |
| Intra-operative failure as assessed by the surgeon | | V | | | |
| Post-operative through Discharge | | $\checkmark$ | le | | |
| Post-operative Repair failure | | | √ | <b>V</b> | V |
| All subjects Pain assessment with VAS | √** | | √** | √** | √* <b>*</b> |
| Satisfaction assessment with VAS | √** | | √** | √** | √** |
| EQ-5D questionnaire | √** | | √** | √** | √** |
| Hip<br>HOOS-ADL score | √** | | √** | √* <b>*</b> | √** |
| Mod. Harris Hip score | √** | | √** | √** | √** |
| Shoulder<br>ROWE Score | √** | | √** | √** | √** |
| ASES score | √** | | √** | √** | √** |
| Constant-Murley score | √** | | √** | √** | √** |
| MRI / Imaging | <b>V</b> | | √* | √* | √* |
| Adverse Event Assessment | | √ | <b>V</b> | | |
| End of Study/Exit | | | √ | | |

<sup>\*</sup> If needed to investigate repair failure

<sup>\*\*</sup> Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

## 3. CONTENTS

## 3.1 TABLE OF CONTENTS

| 1. | Signatures | 2 |
|---|---|---|
| 1.1 | Principal Investigator Signature Page | 2 |
| 1.2 | Sponsor Approval | 3 |
| 2. | Synopsis | 4 |
| 3. | Contents | 10 |
| 3.1 | Table of Contents | 10 |
| 3.2 | Table of Tables | 12 |
| 3.3 | Table of Figures | 12 |
| 3.4 | List of Abbreviations | 13 |
| 4. | Introduction | 16 |
| 4.1 | Background | 16 |
| 4.2 | Literature Summary | 18 |
| 4.3 | Study Purpose | 20 |
| 4.4 | Safety Considerations | 21 |
| 5. | Objective(s) | 22 |
| 5.1 | Primary Objective | 22 |
| 5.2 | Secondary Objective(s) | 22 |
| 6. | Investigational Product(s) | 23 |
| 6.2 | Product Use | 27 |
| 6.3 | Packaging and Labelling | 27 |
| 6.4 | IP/ Ancillary Products and Study Supplies Accountability Procedures | 27 |
| 6.5 | Surgical Technique | 27 |
| 7. | Subject Enrollment and Withdrawal | 28 |
| 7.1 | Subject Population | 28 |
| 7.2 | Inclusion Criteria | 28 |
| 7.3 | Exclusion Criteria | 29 |
| 7.4 | Screening | 30 |
| 7.5 | Informed Consent | 31 |
| 7.6 | Enrollment | 32 |
| 7.7 | Lost to Follow-Up | 32 |

# Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06


| Page: | : Page | 11 | of | 87 |
|-------|--------|----|----|----|

| 7.8 | | Withdrawal | 32 |
|------|-----|-----------------------------------------------------|----|
| 8. | Stu | dy Design | 33 |
| 8.1 | | Study Design | 33 |
| 8.2 | | Allocation and Blinding | 35 |
| 8.3 | | Study Endpoints | 35 |
| 8.4 | | Methods Used to Minimize Bias and Maximize Validity | 36 |
| 9. | Stu | dy Procedures | 37 |
| 9.1 | | Visits and Examinations | 37 |
| 9.2 | | Study Methods and Measurements | 44 |
| 9.3 | | Health Economics/Quality of Life | 44 |
| 10. | Sta | tistical Design | 44 |
| 10. | 1 | General | 45 |
| 10. | 2 | Analysis Populations | 46 |
| 10. | 3 | Baseline Data | 46 |
| 10. | 4 | Efficacy Analysis | 46 |
| 10. | 5 | Safety Analyses | 50 |
| 10. | 6 | Interim Analyses | 50 |
| 11. | Sai | mple Size Justification | 50 |
| 12. | Adv | verse Events and Device Deficiencies | 51 |
| 12. | 1 | Definitions | 51 |
| 12. | 2 | Reporting Procedures | 54 |
| 12. | 3 | Unblinding of Investigational Product | 55 |
| 12. | 4 | Follow-up of Subjects with Adverse Events | 56 |
| 13. | Inv | estigator Obligations | 56 |
| 14. | Spo | onsor and Monitor Responsibilities | 57 |
| 14. | 1 | Contract Research Organization | 57 |
| 14. | 2 | Site Qualification Visit | 57 |
| 14. | 3 | Site Initiation Visit | 57 |
| 14.4 | | Sponsor Audits and Regulatory Inspection | 58 |
| 14. | 5 | Close-out Visit | 58 |
| 15. | Pro | otocol Amendments | 58 |
| 16. | Co | nfidentiality of the Study | 58 |
| 17. | Sta | tements of Compliance | 58 |
| 18. | End | d of Study | 59 |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06


Page: 

| 19. | Pul | blication Policy | 59 |
|---|---|---|---|
| 19 | .1 | Publication of Study Data | 59 |
| 19 | .2 | Data Sharing | 59 |
| 20. | Re | ferences | 60 |
| 21. | App | pendices | 63 |
| 21 | .1 | Instructions For Use Suturefix Ultra and Suturefix curved | 63 |
| 21 | .2 | Protocol Amendment | 66 |
| 21 | .3 | Quality of Life Measures eQ-5D-5L | 67 |
| 21 | .4 | Additional assessments <sup>27</sup> | 69 |
| 21 | .5 | Principal Investigator Obligations (ISO 14155:2011) | 79 |
| 3.2 | T | ABLE OF TABLES | |
| Table | 9.1. | 1-1: Study Procedures by Visit | 37 |
| Table | 12.1 | I-1: Categories of Adverse Event | 51 |
| 3.3 | T | ABLE OF FIGURES | |
| Figur | e 8.1 | -1: Study Flowchart | 34 |
| Figur | <u>- 12</u> | 3-1: Evaluation and Reporting of AE and DevD | 55 |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

## 3.4 LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| ADE | Adverse Device Effect(s) |
| AE | Adverse Event(s) |
| ASES | American Shoulder and Elbow Surgeons Shoulder Score |
| BSI | British Standards Institute |
| CAPA | Corrective and Preventive Action |
| CE | Conformité Européene |
| CI | Confidence Interval |
| CRF | Case Report Form(s) |
| CRO | Contract Research Organization |
| СТ | Computed Tomography |
| СТА | Clinical Trial Agreement |
| CV | Curriculum Vitae |
| DevD | Device Deficiency(ies) |
| EQ-5D | EuroQol 5D |
| FAS | Full Analysis Set Population |
| FDA | Food and Drug Administration |
| FAI | Femoroacetabular Impingement |
| FU | Follow-Up |
| GCP | Good Clinical Practice |
| HIPAA | Health Information Portability Accountability Act |
| HHS | Harris Hip Score |
| HOOS | Hip Disability and Osteoarthritic Outcome Scores |
| HOOS-ADL | Hip Outcome Score Activities of Daily Living |
| IB | Investigator Brochure |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

| Abbreviation | Definition |
|---|---|
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use |
| ICMJE | International Committee of Medical Journal Editors |
| IEC | Independent Ethics Committee |
| IFU | Instructions for Use |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| ISF | Investigator Site File |
| ITT | Intention to Treat population |
| MDI | Multi-directional Instability |
| MITT | Modified Intention-to-treat Population |
| MRI | Magnetic Resonance Imaging |
| NA or N/A | Not Applicable |
| PI | Principal Investigator |
| PP | Per-protocol Population |
| PRO | Subject Report Outcome |
| ROWE | ROWE Shoulder Score for Instability |
| S&N | Smith & Nephew |
| SADE | Serious Adverse Device Effect(s) |
| SAE | Serious Adverse Event(s) |
| SAF | Safety population |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SLAP | Superior Labrum Anterior-Posterior |
| USADE | Unanticipated Serious Adverse Device Effect(s) |

| Suturefix Ultra Suture Anchor Suturefix Curved Suture Anchor | *smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market 1 year Clinical | <b>Number:</b> 17-5010-06 |
| Follow-up Study to evaluate safety and performance of | Version: 1.0, 09/MAY/2018 |
| the SUTUREFIX ULTRA and SUTUREFIX CURVED | <b>Page:</b> Page <b>15</b> of <b>87</b> |
| Suture Anchors in shoulder and hip arthroscopic repair | |

| Abbreviation | Definition |
|--------------|-----------------------|
| VAS | Visual Analogue Scale |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Number:** 17-5010-06

Page: 

### 4. INTRODUCTION

#### 4.1 BACKGROUND

### Shoulder

The superior labrum and biceps anchor improve joint stability by acting like a secondary stabilizer to the shoulder. Labral injuries are usually associated with anterior shoulder dislocation.<sup>1</sup> Diagnosis can be established through MRI by visualizing the distinct line of signal contrast that lies between the glenoid's osseous structure and the glenoid labrum.<sup>1</sup> SLAP (superior labrum anterior-posterior) lesions which were once mainly associated with overhead throwing athletes, are now being diagnosed in older populations.<sup>2</sup> SLAP Lesions are classified into 4 types based on tear stability and location. SLAP tears are a detachment of the superior glenoid labrum from anterior to posterior with or without involvement of the anchor of the long head of the biceps tendon. These tears are typically the result of traction or compression injuries or repetitive overhead activity.<sup>3-5</sup>

Nonoperative treatment such as physical therapy, strengthening programs, antiinflammatories and activity modification, should be considered prior to any surgical intervention. The primary goal of conservative treatment is improvement in shoulder range of motion through posterior capsular flexibility and strengthening of the rotator cuff.<sup>6</sup> When conservative treatment fails to improve symptoms, surgical intervention may be required. Surgical treatments can include simple debridement, stabilization of the biceps-labrum complex through repair, or biceps tenodesis.<sup>7</sup>

Several techniques are utilized for SLAP tear repair, the most common consists of repairing the labrum and biceps anchor.<sup>8</sup> The treatment methods for SLAP repair in younger populations as compared to older populations may vary. Older populations have reported pain and stiffness after SLAP repair.<sup>2</sup> In a systematic review of the literature comparing the treatment in patient over 40 years to patients younger, Erickson et al.<sup>2</sup> found similar outcomes in both populations after SLAP repair.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06

Page: 

Common complications associated with SLAP repair include hardware failure, glenoid osteochondrolysis, and limited range of motion. Hardware failure can include suture anchor pull out, or iatrogenic cartilage damage during instrumentation. Prominent suture knots or hardware have reportedly caused glenoid osteochondrolysis as well<sup>8</sup>. A scarce vascular supply to the superior labrum near the biceps where shear forces are high can contribute to SLAP repair failure as a result of lack of healing.<sup>8</sup>

Outcomes of SLAP repairs have been reported good throughout the literature, with reported success rates ranging from 71-97%, depending on the type of implant used.<sup>3</sup> Patients typically take up to 6 months to regain full motion after SLAP repairs, as stiffness is a common postoperative occurrence, which can be treated with physical therapy and/or subacromial or glenohumeral injections.<sup>3,4,8</sup>

Return to sport is important for many patients with shoulder injuries. Typically the criteria for patients to return to sport include no pain, normal range of motion (ROM), near normal/normal strength, normal functional ability, and patient subjectivity. Usually 14-16 weeks is enough for athletes to return, however it may take as long as 9-12 months. Patients may be hesitant to return to sport for fear of further injury, but those with no restrictive symptoms should be encouraged to return to full activity.

The Constant score, which was developed in 1986, is also rated on a 100-point scale, of which 35 points are based on patient rating. This outcome measure is validated for shoulder arthroplasty, rotator cuff repair, adhesive capsulitis of the shoulder, and proximal humeral fractures. Like the ASES outcome score, higher Constant scores indicate better outcomes. The minimal clinically important difference for this score is not known.<sup>10</sup>

### Hip

The labrum of the hip is a fibrocartilaginous tissue that connects to the osseous edge of the acetabulum, and deepens the acetabular socket while extending coverage of the femoral head. The labrum aids in hip stabilization, by creating negative pressure against distraction and increasing the resistance to dislocation.<sup>11</sup> Femoroacetabular impingement (FAI) is an abnormality of the structure and orientation of the hip joint, which can cause pain and early

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

hip osteoarthrosis.<sup>12-16</sup> Skendzel et al.<sup>15</sup> reported several retrospective reviews which have shown between 49-87% of all patients with a labral tear, have osseous changes consistent with FAI. Chondral injuries have been associated with labral tears and FAI.<sup>17</sup> <sup>15,18</sup> Confirmation of FAI diagnosis usually is achieved with MRI or CT, by reviewing several parameters such as α angle or head-neck offset for cam-type FAI.<sup>11,18</sup> Conservative treatment, such as rest, physiotherapy, and NSAIDs, is usually the first treatment option after FAI diagnosis.<sup>15,18,19</sup> When conservative treatment fails to improve symptoms, surgical intervention may be required. Surgical treatments include debridement, repair and reconstruction, performed either open, arthroscopically, or mini-open.<sup>11,16,18</sup> When labral repair is performed, suture anchors are typically placed onto the acetabular rim, ensuring they do not violate the extra-articular portion of the bone.<sup>16</sup>

The goal of surgical intervention is to restore normal hip mechanics and treating existing damage. Surgical options to treat FAI include Labral debridement and/or repair. <sup>12</sup> <sup>13,15</sup> In an epidemiology study published in 2017, labral pathology was the most common diagnosis at 82% of the population. Of the 1,124 tears reported, 75.3% were repaired, 13.7% were reconstructed and 7.2% were debrided. <sup>20</sup>

In a systematic review performed by Ayeni et al.<sup>12</sup>, arthroscopic management of FAI resulted in postoperative improvements of modified Harris Hip scores that were greater in patients treated with repair as compared to debridement alone. Open management of FAI in the same systematic review<sup>12</sup> reported mixed results, with one study reporting a statistically significant advantage of labral repair over debridement while another study identified reported no differences.

Common complications reported in management of FAI included failures, reoperations, infection and heterotopic bone formation.<sup>12</sup>

### 4.2 LITERATURE SUMMARY

For this literature review, a thorough analysis of the device usage was conducted for the SUTUREFIX ULTRA Suture and SUTUREFIX CURVED Implants equivalent devices currently

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Number: 17-5010-06

Page: 

on the market. Relevant literature was found pertaining to all indications of the SUTUREFIX ULTRA Suture Implant, specifically, shoulder. Good clinical outcomes were reported in the published literature. Improvements in Constant-Murley Scores as well as Flexilevel scale of shoulder function (FLEX-SF) scores were recorded.

In 2015, Agrawal and Pietrzak<sup>21</sup> published the first clinical study with an all-suture anchor. JuggerKnot 1.4 was used for the repair of triple labrum lesions. The mean number of anchors used in the repair was 11.5 (9-19). The study demonstrated improvement in patient outcomes, consistent healing of anchor tunnels, return to activity, and high patient satisfaction. The authors, however, stated that it is unclear whether instability rates will increase with time or there will be detrimental effects of placing more number of anchors in the shoulder. Radiographic results revealed that the JuggerKnot Soft Anchor did not hinder diagnostic imaging, and no instances of subchondral cysts or tunnel expansion were noted. The suture anchor tracts appeared to be healing with fibrous tissue.<sup>22</sup>

Boileau et al<sup>22</sup> reported the use of SUTUREFIX for Bankart repair in 76 patients, although no relevant outcomes were reported.

No complications specific to the use of the SutureFix or Juggerknot device were reported in the published literature. One patient (4.34%) fell and required revision capsular shift and labrum repair. <sup>22</sup>

## Shoulder

Two clinical publications of the shoulder were identified in the literature which followed 76 patients treated with SutureFix and 18 patients treated with Juggerknot. <sup>24</sup> Mean follow up ranged from 14 to 24 months, with a maximum follow up of 24 months.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06

Page: 

Hip

One clinical publication was identified which used the JuggerKnot device in the hip. Matsuda et al., 2015<sup>23</sup> performed a prospective comparative study to compare arthroscopic treatment of global versus focal pincer FAI using a JuggerKnot anchor. The global group consisted of 15 patients (18 hips) and the focal group consisted of 125 patients (129 hips) with a minimum of 2-year follow up. Labral refixation of the posterior rim was performed with a JuggerKnot anchor, it is mentioned that a curved guide was used on occasion, but the number of patients treated with curved devices was not reported.

4.3 STUDY PURPOSE

This is a prospective, multicenter study to evaluate intra-operative, 6 and 12-month safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors for arthroscopic soft tissue repair to meet PMCF requirements for CE Mark and Notified Body (BSI) when used for any of the following indications:

Hip

Acetabular labrum repair/reconstruction

**Shoulder** 

- Capsular stabilization
  - Bankart repair
  - Anterior shoulder instability
  - SLAP lesion repairs
  - Capsular shift or capsulolabral reconstructions
- Rotator cuff tear repairs
- Biceps tenodesis
- Acromioclavicular separation repairs
- Deltoid repairs

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

## 4.4 SAFETY CONSIDERATIONS

The SUTUREFIX ULTRA and SUTUREFIX CURVED Anchor Systems are intended to be used for soft tissue to bone fixation in the Shoulder and Hip. Representative language of the contraindications and potential adverse effects from SUTUREFIX ULTRA and SUTUREFIX CURVED can be found in the IFU. Cleaning and Sterilization Language can be found on the Reusable Surgical Instruments IFU.

Possible Anticipated Adverse Device Effect (ADE) and anticipated Serious Adverse Device Effect (SADE) as reported in the IFU are:

- Mild inflammatory reaction
- Foreign body reaction
- Infection, both deep and superficial
- Allergic reaction
- Loss of fixation or pullout of suture anchors can occur

Investigators shall record adverse events (AEs) and observed device deficiencies, together with an assessment, in the subject's source data. Investigators are responsible for documenting AEs (AE, ADE, SAE, SADE) as described in section 12.1.1 and device deficiencies on the appropriate CRF and submitting them to the Sponsor according to the timelines described here below. At each contact with the subject, the Investigator must seek information on AEs by specific questioning and, as appropriate, by assessment of the subject. AEs must be recorded in standard English medical terminology.

Unresolved AEs should be followed by the Investigator until the events are resolved, the subject is lost to follow-up or through to the end of the study, whichever timing occurs first. Unresolved AEs at the end of the subject's participation will be monitored by the Investigator as part of the site's normal standard of care.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

# 5. OBJECTIVE(S)

#### 5.1 PRIMARY OBJECTIVE

The purpose of this study is to demonstrate the safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in hip and shoulder arthroscopic repair over a time period of 12 months after arthroscopy.

## **5.1.1 Primary Endpoint**

To assess clinical success rate, defined as subjects without signs of failure and/or reintervention at 6 months, as assessed by the surgeon.

## 5.2 SECONDARY OBJECTIVE(S)

## 5.2.1 Secondary Endpoints

To assess safety and performance, supporting the use of SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchor in hip and shoulder arthroscopy repair by measuring:

- Clinical success rate, defined as subjects without signs of failure and/or re-intervention at 12 months, as assessed by the surgeon
- Intra-operative anchor deployment success rate
- Number of anchors pulled out
- Use of additional anchors as a result of intra-operative failure
- Device-related re-intervention
- Safety evaluation at all time points
- Post-operative clinical success rate and performance assessed with subject reported outcomes as follows:

#### All subjects:

Subject pain assessment with VAS at 6 months\* and 12 months\*

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

- Subject satisfaction assessment with VAS at 6 months\* and 12 months\*
- EQ-5D Questionnaire at 6 months\* and 12 months\*

## Hip subjects:

- Hip Outcome Score Activities of Daily Living (HOOS-ADL) at 6 months\* and 12 months\*
- Modified Harris Hip Score (HHS) at 6 months\* and 12 months\*

## Shoulder subjects:

- ROWE Shoulder Scores at 6 months\* and 12 months\*
- ASES Shoulder Scores at 6 months\* and 12 months\*
- Constant-Murley Shoulder Scores at 6 months\* and 12 months\*

## 6. INVESTIGATIONAL PRODUCT(S)

### **6.1.1 Investigational Products**

The SUTUREFIX Anchor is offered in multiple suture configurations including single and double loaded suture options. The delivery system of these anchors enables the suture implant to be placed in the bone in an un- deployed state. During anchor deployment, tension is applied to the repair sutures. The tension applied to the repair sutures, which are threaded through the anchor suture, cause the anchor suture to bunch up. In its deployed state the anchor has a larger nominal diameter than the hole in which it is inserted, locking it into the bone tunnel (Figure 1). The implanted suture anchor construct retains mechanical stability of the soft tissue to bone construct during the healing period. The anchors are available preloaded with either one #2 suture or two #1 sutures.

<sup>\*</sup> Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Number:** 17-5010-06

Page: 

The anchor suture is composed of a single strand of #5 braided, silicone-coated, polyester, non-absorbable suture marketed under the trade name DURABRAID™. The repair suture is comprised of non-absorbable, uncoated ultra-high molecular weight polyethylene (UHMWPE) marketed under the trade name ULTRABRAID™.



Figure 1. SUTUREFIX Implant



Figure 2. SUTUREFIX ULTRA



Figure 3. SUTUREFIX ULTRA DRILL

The SUTUREFIX ULTRA Suture Anchor consists of three components; an all suture based implant preloaded onto a rigid insertion device (Figure 2 and 3), hole preparation and insertion accessory instruments. The Smith & Nephew SUTUREFIX CURVED Suture Anchor utilizes the same anchor as the SUTUREFIX ULTRA (Figure 1), however it comes preassembled to a flexible insertion device (Figure 4 and 5). These devices are provided sterile, for single use only.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 



Figure 4. SUTUREFIX CURVED

Figure 5. SUTUREFIX CURVED DRILL

The instruments included in this file consist of single-use sterile drills (rigid and flexible), as well as reusable drill guides (straight and curved) and obturators (rigid and flexible) (examples seen below in Figures 4 and 5).



Figure 6. Straight obturator and twist drill

Figured 7. Curved Drill Guide

The devices included in this file do not contain any medicinal substances, tissues or blood products.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

> Drill guide, Fishmouth tip, Disposable; Obturator, Blunt, Disposable; 1.9 mm Drill, disposable



Number: 17-5010-06

Version: 1.0, 09/MAY/2018 Page: 

# 6.1.2 IP-Control

72203961

This is the list of study components.

| SUTUREFIX ULTRA Soft Anchors and Instrumentation<br>Systems for Shoulder | | SUTUREFIX ULTRA Soft Anchors and Instrumentation Systems for Hip | |
|---|---|---|---|
| Reference # | Description | Reference # | Description |
| Anchors | | Anchors | |
| 72203852 | SUTUREFIX ULTRA Anchor 1.7 mm S with one<br>Solid Blue (#2) ULTRABRAID' Suture | 72203841 | SUTUREFIX Ultra Anchor 1.7 mm XL with one (#2<br>ULTRABRAID suture (blue) |
| 72203853 | SUTUREFIX ULTRA Anchor 1.7 mm S with one<br>Blue COBRAID (#2) ULTRABRAID Suture | 72203842 | SUTUREFIX Ultra Anchor 1.7 mm XL with one (#2<br>ULTRABRAID suture (blue-COBRAID) |
| 72203854 | SUTUREFIX ULTRA Anchor 1.9 mm S with two<br>Blue, Blue COBRAID (#1) ULTRABRAID Sutures | <b>Drills</b> 72203843 | SUTUREFIX Ultra Drill 1.7mm XL, Disposable |
| Drills | | | |
| 72203855 | Twist drill 1.7 mm S | Guides & Obture | ators |
| 72203856 | Twist drill 1.9 mm S | 72203844<br>72203845 | Drill Guide XL, Crown Tip<br>Drill Guide XL, Spike Tip |
| Guides & Obtur | rators | 72203846 | Obturator XL, Blunt tip |
| 72203857<br>72203858 | Drill Guide crown tip, Reusable, S<br>Drill Guide Spike tip, Reusable, S | 72203899 | Obturator XL, Cannulated, Blunt Tip |
| 72203859 | Drill Guide Fishmouth tip, Reusable, S | Knot Pusher | |
| 72203861 | Obturator, Blunt tip, Reusable, S | 72203850 | ELITE' Knot Pusher XL |
| 72203862 | Obturator, Cannulated, Reusable, S | | *************************************** |
| 72203863 | Obturator, Trocar tip, Reusable, S | | |
| Anchor Packs | | _ | |
| 72203953 | SUTUREFIX Ultra Anchor S, Box of 3 with one Drill 1.7 mm, Disposable | | |
| 72203954 | SUTUREFIX Ultra Anchor S, Box of 3 with one<br>Drill 1.9 mm, Disposable | | |
| 72203955 | SUTUREFIX Ultra Anchor 1.7 mm S, Box of five | | |
| 72203956 | SUTUREFIX Ultra Anchor 1.9 mm S, Box of five | | |
| Instrumentation | Kits | | |
| 72203957 | Drill guide, Crown tip, Disposable; Obturator,<br>Blunt, Disposable; 1.7 mm Drill, disposable | | |
| 72203958 | Drill guide, <u>Fishmouth</u> tip, Disposable; Obturator,<br>Blunt, Disposable; 1.7 mm Drill, disposable | | |
| 72203959 | Drill guide, <u>Spiked</u> tip, Disposable; Obturator,<br>Blunt, Disposable; 1.7 mm Drill, disposable | | |
| 72203960 | Drill guide, Crown tip, Disposable; Obturator,<br>Blunt, Disposable; 1.9 mm Drill, disposable | | |

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




**Page:** 

## 6.1.3 Ancillary Products

No ancillary products are to be provided.

## 6.2 PRODUCT USE

SUTUREFIX ULTRA and CURVED Suture Anchors are intended for the secure fixation of soft tissue to bone and should be used according to IFU. The non-absorbable suture will remain in the tissue permanently.

Surgeons selected to participate in this study will be experienced with implanting SUTUREFIX ULTRA Suture Anchor and SUTUREFIX CURVED Suture Anchor and no additional training is required.

### 6.3 PACKAGING AND LABELLING

Packaging and labelling will be prepared to meet regulatory requirements.

Commercial products are being used and the standard device procurement and management will be used per site process.

Packaging integrity needs to be confirmed prior to surgery and recorded in the CRF.

#### 6.4 IP/ Ancillary Products and Study Supplies Accountability Procedures

This is a post-market follow-up study. Only commercial available devices are implanted by the hospitals or clinics. All products received regulatory clearance in the countries where the study takes place. Therefore no device accountability is applicable.

### 6.5 SURGICAL TECHNIQUE

All study related procedures with the SUTUREFIX Ultra Suture Anchor and SUTUREFIX Curved Suture Anchor must be performed according to the recommended surgical technique described

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

in the protocol or in a separate instructional document and product labelling (e.g. IFU and package insert) as applicable.

### 7. SUBJECT ENROLLMENT AND WITHDRAWAL

## 7.1 SUBJECT POPULATION

In this study a minimum of 80 subjects will be enrolled, 40 subjects for each group, hip and shoulder. The subjects will be treated with the study device(s) for hip or shoulder instability.

### 7.2 INCLUSION CRITERIA

Subjects will be considered qualified for enrollment if they meet the following criteria:

- 1. Subject has consented to participate in the study by signing the EC-approved informed consent form
- 2. Subject is 18 years of age at time of surgery.
- Subject condition meets proposed indication to SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchor
- 4. Subject requiring shoulder or hip arthroscopic labral repair surgery from physical findings, subject symptoms and radiographic finding
- 5. Bone quality and quantity must be adequate to allow proper placement of the anchor
- 6. Able to follow instructions.
- Willing and able to make all required study visits.

### Hip subjects

8. FAI (Femoroacetabular Impingement)

## **Shoulder subjects**

9. Subject with a history of recurrent dislocation/subluxation of the shoulder

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Number:** 17-5010-06


Page: 

## 7.3 EXCLUSION CRITERIA

Any one (1) of the following criteria will disqualify a potential subject from participation in the study:

## All subjects

- 1. Participation in the treatment period of another clinical trial within thirty (30) days of Visit 1 (pre-operative)
- Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures
- 3. Any subject that meets the definition of a Vulnerable Subject per ISO14155:2011: individual whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate
- 4. Subjects with a history of poor compliance with medical treatment
- Contraindications or hypersensitivity to the use of the SUTUREFIX ULTRA and/or SUTUREFIX CURVED Suture Anchor, or their components (e.g. silicone, polyester). Where material sensitivity is suspected, appropriate tests should be performed and sensitivity ruled out prior to implantation
- 6. Prior ipsilateral surgeries performed on the joint space

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

8. Pathological conditions of bone, such as cystic changes or severe osteopenia, which would compromise secure anchor fixation

- 9. Pathological conditions in the soft tissues to be attached that would impair secure fixation by suture
- 10. Comminuted bone surface, which would compromise secure anchor fixation Physical conditions which would eliminate, or tend to eliminate, adequate anchor support in impair healing
- 11. Epileptic history

## **Hip subjects**

12. Dysplasia latera/central less than 20°

## **Shoulder subjects**

- 13. Glenoid and/or humeral bone loss considered excessive by the treating orthopaedic surgeon
- 14. MDI: Multi-directional instability
- 15. Psychosomatic voluntary shoulder subluxation

#### 7.4 SCREENING

To eliminate the potential for selection bias, Investigators should consecutively pre-screen all subjects undergoing arthroscopic instability repair with SUTUREFIX ULTRA Suture Anchor and/or SUTUREFIX CURVED Suture Anchor. Subjects receiving care at the investigative sites will be pre-screened as potential subjects for the study. To do so, only the existing information obtained per standard routine medical procedures will be used. No study-specific screening procedures, activities or questionnaires will be performed during pre-screening.

Participating study sites are required to document all screened subjects considered for inclusion in this study. If a subject is excluded from the study, the reasons for exclusion will be documented in the subject's source documents and noted on the Screening and Enrollment Log.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

Once a subject has completed the informed consent procedure and signed an Ethics Committee approved Informed Consent Form (ICF), the PI or delegated study research staff can complete the screening process with the subject (see Section 9.1).

All screening activities which occur prior to consent shall be referred to as pre-screening.

#### 7.5 INFORMED CONSENT

Before conducting any study procedures or examinations, the purpose and nature of the study will be explained to the subject in their native language. The ICF will be translated from English master ICF and/or adjusted to the EC requirements to the national languages of the participating European countries. The subject, or their legally authorized representative, will then **read**, **sign**, and **personally date** the IRB/IEC-approved informed consent document(s) (see below for difficulties with reading and writing). Additionally, the individual who obtains consent from the subject will sign and date the informed consent document. A copy of the signed informed consent documentation will be provided to the subject, a copy will be placed in the subject's medical record, with the original filed in the ISF.

If the subject is unable to read, the informed consent document and associated study information may be read aloud to the subject in the presence of an impartial witness. If possible the subject shall sign and personally date the Informed Consent Form (ICF). Where this is not possible, due to difficulties in writing, the subject shall provide verbal consent to participate in the study. The witness shall then personally sign and date the informed consent form, attesting that the information was accurately explained and that the informed consent was freely given.

For the site(s) in United States the HIPPA requirements will be in place.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06

Page: 

#### 7.6 ENROLLMENT

Once a subject has completed the informed consent procedure and signed an Ethics Committee approved Informed Consent Form (ICF) the PI or delegated study research staff can complete the screening process with the subject.

### 7.7 LOST TO FOLLOW-UP

Some actively enrolled subjects will not return for follow-up exams on time. Study personnel must make a reasonable effort to contact the subject and document the following contact attempts prior to declaring a subject to be lost to follow-up: the subject has been contacted according to the site's policies, but no fewer than 2 documented phone contacts and 1 certified letter without response. Copies of all attempts to reach the subjects per regular mail or email and/or the attempts to contact the subject via other means should be documented and that documentation should be kept with the subject's source documents.

### 7.8 WITHDRAWAL

#### 7.8.1 Withdrawal from Treatment

Not applicable

### 7.8.2 Withdrawal from Study

The Investigator **may** withdraw subjects from the study for many reasons, including but not limited to the following:

- subject noncompliance (e.g. did not follow instructions)
- subject lost to follow-up
- if the Investigator or the Sponsor stops the study for any reason and decides to withdraw subject(s) from the study
- Adverse Events/

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

· any other significant reason identified by the Investigator

For each case, information will be obtained in the source document and the Case Report Form (CRF) detailing circumstances leading to the withdrawal.

Subjects who drop out or are withdrawn will not be re-entered into the study at a later date.

## 7.8.3 Subject's Withdrawal of Consent to Participate in Study

Study participation is voluntary and subjects may withdraw at any point during the study without giving their reason for doing so. Where subjects withdraw consent, the Investigator should make a reasonable effort to ascertain the reason(s), while fully respecting the subject's privacy. The reason for withdrawal will be recorded in the CRF and in source documents.

## 7.8.4 Use of Data Following Withdrawal

In cases where the subject withdraws consent, the data collected up to the point of withdrawal may be used but no additional data for that subject may be collected.

#### 8. STUDY DESIGN

#### 8.1 STUDY DESIGN

This is a prospective, multicenter study to evaluate the clinical and intraoperative outcomes from 80 subjects implanted with the SUTUREFIX ULTRA and/or SUTUREFIX CURVED Suture Anchors in hip or shoulder groups. Up to 8 sites (up to 4 sites for study hip group and up to 4 sites for study shoulder group) in Europe will participate in the study. Data from eligible subjects, who have provided written and informed consent for the collection of their coded data (see section 9.1.2-9.1.6) will be recorded from the subject medical file on Case Report Forms (CRFs). Follow-up clinical assessments will be performed at 6 months and 1 year post-operatively.

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06

**Version:** 1.0, 09/MAY/2018 **Page:** 

This is an open-label study with consecutive enrollment. The study will continue for 12 months from the date of treatment for the last subject completing the study as planned. Only subjects who meet the enrollment criteria as listed in section 7 will be enrolled into the study. The study duration is planned for 24 months.

The data will support CE Mark certification for the Shoulder and Hip repair indications. The data should confirm safety and performance levels acceptable for the risk benefit profile of this device.

Pre-Screening Screening **Enrollment and Study Conduct** Verification of eligibility criteria Document subject on screening and per standard routine medical yes enrollment log procedure: Subject eligible? no Complete Informed Consent Procedure yes Perform Assessment 1: Pre-operative Subject willing to participate? visit and complete pre-operative CRFs No further action Update screening and enrollment log. No Perform Assessment 2: Surgery and CRFs will be collected complete intra-operative and discharge **CRFs** Perform Assessment 3: 6-months followup visit and complete CRFs Perform Assessment 4: 12-months follow-up call and complete CRFs

Figure 8.1-1: Study Flowchart

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

### 8.2 ALLOCATION AND BLINDING

This study is an open-label study with consecutive enrolment without randomization. There is no control group. Although there are two groups one hip and one shoulder group blinding of the surgeon is not applicable due to the different indications and product specificities. The evaluator will be blinded to the treatment groups.

### 8.3 STUDY ENDPOINTS

## 8.3.1 Primary Endpoint

 Clinical success rate, defined as subjects without signs of failure and/or re-intervention at 6 months, as assessed by the surgeon

## 8.3.2 Secondary Endpoints

- Clinical success rate, defined as subjects without signs of failure and/or re-intervention at 12 months, as assessed by the surgeon
- Intra-operative anchor deployment success rate
- Number of anchors pulled out
- Use of additional anchors as a result of intra-operative failure
- Device-related re-intervention
- Safety evaluation at all time points
- Post-operative clinical success rate and performance assessed with subject reported outcomes as follows:

# All subjects:

- Subject pain assessment with VAS at 6 months\* and 12 months\*
- Subject satisfaction assessment with VAS at 6 months\* and 12 months\*
- EQ-5D Questionnaire at 6 months\* and 12 months\*

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

# Hip subjects:

- Hip Outcome Score Activities of Daily Living (HOOS-ADL) at 6 months\* and 12 months\*
- Modified Harris Hip Score (HHS) at 6 months\* and 12 months\*

### Shoulder subjects:

- ROWE Shoulder Scores at 6 months\* and 12 months\*
- ASES Shoulder Scores at 6 months\* and 12 months\*
- Constant-Murley Shoulder Scores at 6 months\* and 12 months\*

### 8.4 METHODS USED TO MINIMIZE BIAS AND MAXIMIZE VALIDITY

The study is a prospective multi-centre non-comparative cohort study to demonstrate the performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in hip and shoulder for arthroscopic treatment over a time period of 12 months after arthroscopy. The study is exploratory in nature and not powered for any statistical testing hence the results from the study will be interpreted with caution.

Biases naturally associated with exploratory non-comparative studies will be inevitable but the use of multiple recruitment centres and well defined inclusion/exclusion criteria ensures that the study is more representative of a larger population and varying backgrounds. The exploratory data analysis planned for the study which includes confidence intervals for the outcome summaries, a pre-defined confidence interval for the primary outcome and exploratory statistical models adjusting for potential confounding factors is designed to maximise the validity of the study results.

<sup>\*</sup> Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference
## Suturefix Ultra Suture Anchor Suturefix Curved Suture Anchor

Prospective, Multicenter, Post-Market 1 year Clinical Follow-up Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Number:** 17-5010-06

**Version:** 1.0, 09/MAY/2018 **Page:** 

### 9. STUDY PROCEDURES

#### 9.1 VISITS AND EXAMINATIONS

#### 9.1.1 Summary

For a summary of the required procedures by visit, refer to Table 9.1-1: Study Procedures by Visit

Table 9.1.1-1: Study Procedures by Visit

| Cohodula of sucreta (top recoded) | Visit 1 | Visit 2 | Visit 3<br>Visit | Visit 4 Telephone Call or Visit | Visit 5<br>Unscheduled<br>Visit |
|---|---|---|---|---|---|
| Schedule of events (*as needed) | Pre-<br>Operative | Operative<br>through<br>Discharge | 6 Months<br>(± 1 M) | 12 Months<br>(± 1 M) | |
| Informed Consent | V | | | | |
| Inclusion/Exclusion Criteria | V | | | | |
| Demographics/ Medical History | $\checkmark$ | | | | |
| Intra-op failure as assessed by the surgeon | | <b>√</b> | | | |
| Operative through Discharge | | $\sqrt{}$ | | | |
| Post-op Repair failure | | | √ | <b>√</b> | $\checkmark$ |
| All subjects Pain assessment with VAS | √** | | √** | √** | √** |
| Satisfaction assessment with VAS | √** | | √** | √** | √** |
| EQ-5D questionnaire | √** | | √** | √** | √** |
| Hip<br>HOOS-ADL score | √** | | √** | √** | √** |
| Mod. Harris Hip score | √** | | √** | √** | √** |
| Shoulder<br>ROWE score | √** | | √** | √** | √** |
| ASES score | √** | | √** | √** | √** |

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06

**Version:** 0.17, 17/APR/2018

Page: 

| Cabadula of avents (tag panded) | Visit 1 | Visit 2 | Visit 3<br>Visit | Visit 4 Telephone Call or Visit | Visit 5<br>Unscheduled<br>Visit |
|---|---|---|---|---|---|
| Schedule of events (*as needed) | Pre-<br>Operative | Operative<br>through<br>Discharge | 6 Months<br>(± 1 M) | 12 Months<br>(± 1 M) | |
| Constant-Murley score | √** | | √** | √** | √** |
| MRI / Imaging | √ | | √* | √* | √* |
| Adverse Event Assessment | | V | $\sqrt{}$ | | |
| End of Study/Exit | | | √ | | |

<sup>\*</sup> If needed to investigate repair failure

<sup>\*\*</sup> Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06 Version: 1.0, 09/MAY/2018 Page: 

#### 9.1.2 Visit 1: Pre-Operative Visit

Obtain written informed consent from the subject as detailed in Section 7.5

#### ---- Do not proceed until consent has been obtained ----

- Obtain demographic information and medical history, including information on all concomitant medications/therapies
- Screen the subject for protocol inclusion/exclusion criteria
- Assign the subject a study number and instruct the subject on treatment procedures
- Complete Screening and Enrollment Log
- Complete VAS-Scale for Pain for all subjects\*
- Complete EQ-5D questionnaire for all subjects\*
- Complete ROWE Score for shoulder\*
- ASES Score for shoulder\*
- Complete Constant-Murley Score for shoulder\*
- Complete HOOS-ADE Score for hip\*
- Complete Modified HSS Sore for hip\*
- Perform MRI, only in case of repair failure
- If any adverse events are observed or reported, they must be recorded as instructed in Section 12.3, adverse events and device deficiencies
- Complete Pre-Operative Visit CRFs

<sup>\*</sup>Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06 Version: 1.0, 09/MAY/2018

Page: 

#### 9.1.3 Visit 2: Operation through Discharge Visit

- Query subject regarding any changes in general health and the use of concomitant medications
- If any adverse device effects or device deficiencies are observed or reported, they
  must be recorded as instructed in Section 12.3 adverse events and device
  deficiencies
- Update information in the Screening and Enrollment Log
- Intra-operative success as assessed by the surgeon
- MRI/Images, only in case of repair failure
- Complete Operation and Discharge Visit CRFs
- Instruct the subject on follow-up procedures, including returning to the facility for FU
   Visit 3 in (± 1M) 6 months

#### 9.1.4 Visit 3: 6-Month Follow-up Visit (± 1 month)

- Query subject regarding any changes in general health and the use of concomitant medications.
- If any adverse device effects or device deficiencies are observed or reported, they
  must be recorded as instructed in Section 12.3, adverse events and device
  deficiencies
- Post-operative repair failure
- Complete VAS-Scale for Pain and Satisfaction for all subjects\*
- Complete EQ-5D questionnaire for all subjects\*
- Complete ROWE Score for shoulder\*
- ASES Score for shoulder\*
- Complete Constant-Murley Score for shoulder\*
- Complete HOOS-ADE Score for hip\*

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

| 'emith | 2.no | ahaw |
|--------|-------|------|
| smith | ionie | |


**Page:** 

- Complete Modified HSS Sore for hip\*
- · Perform MRI/Imaging only in case of repair failure
- Complete 6-Months Follow-up Visit CRFs
- Instruct the subject on follow-up procedures, including scheduling a FU call or visit in (± 1M) 12 months

\*Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference.

#### 9.1.5 Visit 4: 12-Months Follow-up Call or Visit (± 1 month)

- Query subject regarding any changes in general health and the use of concomitant medications.
- If any adverse device effects or device deficiencies are observed or reported, they
  must be recorded as instructed in Section 12.3, adverse events and device
  deficiencies.
- Post-operative repair failure
- Complete VAS-Scale for Pain and Satisfaction for all subjects\*
- Complete EQ-5D questionnaire for all subjects\*
- Complete ROWE Score for shoulder\*
- ASES Score for shoulder\*
- Complete Constant-Murley Score for shoulder\*
- Complete HOOS-ADE Score for hip\*
- Complete Modified HSS Sore for hip\*
- Perform MRI/Imaging only in case of repair failure

\*Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06 Version: 1.0, 09/MAY/2018

**Page:** 

#### 9.1.6 Unscheduled Visits

- Query subject regarding any changes in general health and the use of concomitant medications.
- Adverse device effects or device deficiencies must be recorded as instructed in Section 12.3, adverse events and device deficiencies.
  - Post-operative repair failure
- Complete VAS-Scale for Pain and Satisfaction for all subjects\*
- Complete EQ-5D questionnaire for all subjects\*
- Complete ROWE Score for shoulder\*
- ASES Score for shoulder\*
- Complete Constant-Murley Score for shoulder\*
- Complete HOOS-ADE Score for hip\*
- Complete Modified HSS Sore for hip\*
- Perform MRI/Imaging to investigate repair failure
- Complete Unscheduled Visit CRFs
  - \*Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference

Unscheduled examinations may be conducted at the discretion of the Investigator with all obtained information recorded in the source documents and on the appropriate CRF.

#### 9.1.7 Concomitant Medications and Therapies

A concomitant medication (e.g. drug, substance) and a concomitant therapy (e.g. physical therapy, TENS Unit, massage) are recorded at any time from enrollment into the study through the subject's last study visit.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06 Version: 1.0, 09/MAY/2018

Page: 

#### 9.1.7.1 Concomitant Medications

#### **9.1.7.1.1** Excluded Concomitant Medications

Not applicable

#### **9.1.7.1.2** Recording Concomitant Medications in the CRF

Concomitant medications should be recorded in the CRF with the generic name.

#### 9.1.7.2 Concomitant Therapies

#### **9.1.7.2.1** Therapies Prohibited During the Study

Not applicable

#### 9.1.7.2.2 Recording Concomitant Therapies in the CRF

Standard concomitant therapy will be recorded in the CRF unless provided as a part of an AE treatment.

#### 9.1.8 Discontinued Subjects

Discontinued subjects are those who voluntarily discontinue participation, who are withdrawn for reasons of safety, who are lost to follow-up, so are ineligible for further participation, refer to section 7.8 for further details. Where possible, a full Exit Visit should be completed for all subjects who discontinue the study early. Where consent is withdrawn, the date and any reason given for discontinuation should be captured, at a minimum (see Section 7.8.2).

Finally, if appropriate, the Investigator will also advise the subject of subsequent therapy and/or procedures necessary for their medical condition.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair smith&nephew


Page: 

#### 9.1.9 Subject Pregnancy

Women of child-bearing potential are not excluded from the study: as long as adequate birth control methods are being used by the subject as outlined in the protocol's exclusion criteria. However, if a woman becomes pregnant during the study, S&N must be contacted immediately once the investigator is made aware of the pregnancy and a decision will be made regarding the continuation in the study of the pregnant woman. Pregnancy is not an adverse event; however, complications related to the pregnancy may be reportable as determined on a case-by-case basis. Pregnancy-related information will be collected until the end of the pregnancy.

#### 9.2 STUDY METHODS AND MEASUREMENTS

#### All subjects

VAS for pain and satisfaction assessment\*

#### Hip subjects

- Hip Outcome Score Activities of Daily Living (HOOS-ADL)\*
- Modified Harris Hip Score (HHS) \*

#### **Shoulder subjects**

- ROWE Shoulder Scores\*
- ASES Shoulder Scores\*
- Constant-Murley Shoulder Scores\*

\*Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference

#### 9.3 HEALTH ECONOMICS/QUALITY OF LIFE

• EQ-5D-5L

#### 10. STATISTICAL DESIGN

The primary aim of the study is to evaluate intra-operative (6 and 12-month) safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors for arthroscopic repair. This section of the protocol is a brief description of the analyses projected to

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair smith&nephew


Number: 17-5010-06

Page: 

evaluate the aims of the study and answering the study research question. A more detailed Statistical Analysis Plan (SAP) will be written and finalized prior to database lock. The SAP will account for any changes or deviations from the projected analyses in this protocol.

#### 10.1 GENERAL

Primary and secondary endpoints will be evaluated using listings and appropriate summary statistics. The outcomes will be summarized for the entire sample, by device implanted (SUTUREFIX ULTRA and SUTUREFIX CURVED) as well as the position, i.e. the hip or the shoulder. The summary statistics for both primary and secondary outcomes will be reported together with a 95% confidence interval where necessary to assess the degree of precision in the estimates.

Data tabulations and summarization will be presented to aid in the interpretation of the effects of clinically important variables that are disclosed. A summary of the enrolment figures by site, time point follow-up as well as the demographic and baseline variables, which include age, gender etc. will be presented. Continuous variables will be summarized using mean, median, SD, minimum, and maximum; categorical variables will be summarized as counts and percentages.

All statistical tests will be exploratory in nature as the study is not powered for any statistical testing. Appropriate parametric and/or non-parametric analyses will be chosen for statistical analysis. Test of association for the table of counts will be based on the Fisher's Exact Test unless otherwise inappropriate. The exploratory analysis of continuous variables will be done using t-test and ANOVA if appropriate. The Wilcoxon rank-sum or Kruskal-Wallis tests will be explored if the data is non-normal.

For the success/failure variable, the logistic model will be considered if needed. Associated factors will be adjusted for in unadjusted and adjusted models, if necessary (Peacock and Kerry 2007).<sup>25</sup> All statistical tests and models will be considered at 5% significance level. Adverse Events will be tabulated for the study duration.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06


**Page:** 

All statistical analyses and calculation of confidence intervals will be performed using SAS software.

#### 10.2 ANALYSIS POPULATIONS

All subjects who provide informed consent are considered study participants. Study populations are defined as follows:

- Full analysis set population (FAS), including all subjects who were enrolled into the study and attended at least one post-baseline assessment.
- Per-Protocol Population (PP), including all subjects in the full analysis set who have no significant protocol deviations and met the inclusion/exclusion criteria.
- Safety Population (SAF), including all subjects who have received IP.

#### 10.3 BASELINE DATA

Data to be summarised at baseline includes all collected demographic variable such as age, gender, primary diagnosis, height, weight, BMI, medical history and co-morbid conditions. The baseline variables will be used to describe the outcome data where necessary. Continuous baseline data will be summarized using frequency, means, and standard deviations, median, minimum and maximum. Categorical variables will be summarized using counts and percentages. The percentages will be calculated based on the number of non-missing values.

#### 10.4 EFFICACY ANALYSIS

#### **10.4.1 Analysis of Primary Endpoint**

Clinical success rate, defined as subjects without a signs of failure and/or re-intervention at 6 months, surgeon assessment:

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair \*smith&nephew


Page: 

• The frequency of the subjects without a signs of failure and/or re-intervention at 6 months together with percentage with a 95% CI will be reported. Clinical success rate for the entire sample, by device implanted (SUTUREFIX ULTRA and SUTUREFIX CURVED) as well as the position, i.e. the hip or the shoulder will be reported. A binary variable of success/failure will be used to fit a logistic model adjusting device implanted and position to estimate the odds ratio of success if data allows.

#### 10.4.2 Analysis of Secondary Endpoint(s)

- Intra-operative anchor deployment success rate
- Number of anchors pulled out
- Use of additional anchors as a result of intra operative failure
- Device-related re-intervention

All the above variables will be categorical in nature hence frequencies together with percentages will be tabulated for the entire sample as well as by device implanted (SUTUREFIX ULTRA and SUTUREFIX CURVED) as well as the position, i.e. the hip or the shoulder will be reported.

#### All subjects

Clinical success rate, defined as subjects without signs of failure and/or re-intervention at 12 months; surgeon assessment

- The frequency of the subjects without a signs of failure and/or re-intervention at 12 months together with percentage with a 95% CI will be reported. Clinical success rate for the entire sample, by device implanted (SUTUREFIX ULTRA and SUTUREFIX CURVED) as well as the position, i.e. the hip or the shoulder will be reported. A binary variable of success/failure will be used to fit a logistic model adjusting device implanted and position to estimate the odds ratio of success if data allows.
- Subject pain assessed with a VAS at 6 months\* and 12 months\*

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

Subject satisfaction assessed with a VAS at 6 months\* and 12 months\*

EQ-5D Questionnaire at 6 months\* and 12 months\*

The VAS and EQ-5D-5L scores at different time points and end of study for the entire sample, by device implanted (SUTUREFIX ULTRA and SUTUREFIX CURVED) as well as the position, i.e. the hip or the shoulder will be summarized using mean, median, SD, minimum, and maximum. A one sample t-test will be used to test the difference between baseline and end of study scores. A non-parametric test will be considered if necessary.

#### • EQ-5D-5L

Based on the subjects responses (no problems/some or moderate problems/extreme problems) to each dimension (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) an index utility score is calculated to represent the overall EQ-5D-5L score for each subject.

The subject responses to each dimension score and the overall EQ-5D-5L index utility scores and EQ VAS scores will be summarized at baseline and all post-operative visits for the entire sample, by device type implanted and as well as the position, i.e. the hip or the shoulder.. The change in EQ-5D-5L index utility score and the change in EQ VAS score between baseline and all post-op visits will also be summarised.

EQ-5D-5L Utility scores and EQ VAS scores will be assessed using separate repeated measures ANOVA model, with the relevant score as the dependent variable for on entire sample with device implanted and position accounted for as levels in the model.

#### Hip subjects

 Hip Outcome Score Activities of Daily Living (HOOS-ADL) at 6 months\* and 12 months\*

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06 Version: 1.0, 09/MAY/2018

**Page:** 

Modified Harris Hip Score (HHS) at 6 months\* and 12 months\*

The HOOS and HHS scores at different time points and end of study will be will be summarized for the entire sample and device implanted using median, SD, minimum, and maximum. A one sample t-test will be used to test the difference between baseline and end of study scores.

#### **Shoulder subjects**

- ROWE Shoulder Scores at 6 months\* and 12 months\*
- ASES Shoulder Scores at 6 months\* and 12 months\*
- Complete Constant-Murley Score for shoulder\* at 6 months\* and 12 months\*
  - The ROWE and Constant-Murley Shoulder scores at different time points and end of study will be will be summarized for the entire sample and device implanted using mean, median, SD, minimum, and maximum. A one sample t-test will be used to test the difference between baseline and end of study scores. A nonparametric test will be considered if necessary.

\*Patient Reported Outcomes (PROs) are optional and used according to the surgeon's preference

#### 10.4.3 Analysis of Other Endpoint(s)

Time to failure - intra-operative repair failure will be defined as just an event.

- If adequate data is available, Kaplan Meier survival estimate for the entire sample, by device implanted and position will be used in this study survival analyses and a Cox model will also be explored adjusting for device implanted and position.
- Available data will be summarized and summary statistics tabulated.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06
Page: 

#### 10.5 SAFETY ANALYSES

Adverse events

 Adverse Events (as defined in Safety Reporting Section – All adverse events will be tabulated classified by seriousness and given by frequency and percentages for the entire sample and by device implanted (SUTUREFIX ULTRA and SUTUREFIX CURVED).

#### 10.6 INTERIM ANALYSES

No interim analysis is foreseen.

#### 11. SAMPLE SIZE JUSTIFICATION

A systematic review by Erickson et al (2015) suggests that the variation in the success rate among patients who have undergone any Suture Anchors for arthroscopic instability repair range from 71-97%. Two studies Lafosse et al (2008) and Thal et al (2007) <sup>26</sup> have failure rates of 11.4% and 6.9% within a period of 2 years from surgery, giving success rates of about 87% and 93% respectively suggest that building a 11% confidence interval either side of 89% will ensure that the estimated success rate is within literature extrapolated success rates.

This study considers the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors for arthroscopic repair success rate and a sample of 80 (40 per device) subjects is considered. A sample size of 40 subjects will estimate a success rate of 89% with a 95% confidence interval (CI) [78: 100] with 55% probability.

| Study Protocol—Device | %smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market Clinical Follow- | Number: 17-5010-06 |
| up Study to evaluate safety and performance of the | Version: 1.0, 09/MAY/2018 |
| SUTUREFIX ULTRA and SUTUREFIX CURVED Suture | Page: |
| Anchors in shoulder and hip arthroscopic repair | |

#### 12. ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 12.1 **DEFINITIONS**

The categories of adverse events are shown in table 12.1-1. The definitions for each of these categories are given in the subsequent sections (see reference within the table).

**Table 12.1-1: Categories of Adverse Event** 

| | NOT DEVICE-<br>RELATED | DEVICE- OR PROCEDURE-RELATED | |
|---|---|---|---|
| NON-<br>SERIOUS | ADVERSE EVENT (AE) (SEE 12.1.1) | Adverse Device Effect<br>(ADE) (see 12.1.2) | |
| | Serious Adverse | Serious Adverse Device Effect<br>(SADE) (see 12.1.3) | |
| SERIOUS | EVENT | ANTICIPATED | UNANTICIPATED |
| <b>32</b> 141 <b>333</b> | (SAE)<br>(SEE 12.1.3) | ANTICIPATED SERIOUS<br>ADVERSE DEVICE EFFECT<br>(ASADE) (SEE 12.1.4) | UNANTICIPATED SERIOUS<br>ADVERSE DEVICE EFFECT<br>(USADE) (SEE 12.1.4) |

#### 12.1.1 Adverse Event

An <u>Adverse Event (AE)</u> is any untoward medical occurrence between enrollment (signed ICF obtained) and study discontinuation with the use of an IP, whether or not considered causally related to that IP.

AE is used both to refer to AE which are non-serious non-IP or procedure-related and as an umbrella term referring to adverse events of all classifications.

An AE can be any unfavorable and unintended sign (for example, an abnormal laboratory finding), symptom, or disease. For reporting purposes, emphasis is placed first and foremost on whether or not the event constitutes an <u>untoward medical occurrence</u>.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06 Version: 1.0, 09/MAY/2018

**Page:** 

#### 12.1.2 Adverse Device Effect

An <u>Adverse Device Effect (ADE)</u> is an adverse event that, in the opinion of the investigator, is related to the IP or the procedure.

Not Related - An AE is considered to be not related to the use of an IP or the procedure when the effect is DEFINITELY UNRELATED or UNLIKELY to have any relationship to the use of the IP or the procedure;

**Related** - An AE is considered to be related to the use of an IP or the procedure when there is a POSSIBLE, PROBABLE, or DEFINITE relationship between the AE and the use of the IP or the procedure.

An ADE is further categorized depending on whether the criteria in section 12.1.3 and 12.1.4 are met.

#### 12.1.3 Serious Adverse Events and Serious Adverse Device Effects

An AE or ADE is considered a **Serious** Adverse Event (SAE) or **Serious** Adverse Device Effects (SADE) if, in the view of either the Investigator or the Sponsor, it:

- Results in death.
- Is life-threatening (*NOTE*: The term "life-threatening" in the definition of "serious" refers to an event/reaction in which the subject was at risk of death at the time of the event/reaction; it does not refer to an event/ reaction which hypothetically might have caused death if it were more severe).
- Requires in subject hospitalization or results in prolongation of existing hospitalization.
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- Is a congenital anomaly/birth defect.
- Is a medically important event or reaction.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious such as important medical events that might not be immediately life-threatening or result in death or hospitalization but might jeopardize the subject or might require intervention to prevent one of the other outcomes listed in the definition above. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse.

#### 12.1.4 Anticipated/Unanticipated Serious Adverse Device Effect

An Unanticipated Serious Adverse Device Effect (USADE) is a serious ADE that meets any of the above definitions but is also considered, by the Investigator, to be caused by or related to the IP, not previously identified in nature, severity or degree in the IFU <sup>28,29,30</sup>.

An Anticipated Serious Adverse Device Effect (ASADE) is a serious ADE that does not meet the criteria for a USADE <sup>28,29,30</sup>.

#### 12.1.5 Severity

The severity of every AE will be assessed by the PI or medically qualified site staff to whom the responsibility has been delegated and documented on the delegation of authority log. AE should be classified as mild, moderate, or severe, regardless of whether or not the AE are considered to be serious or non-serious. The classification should be based on the following definitions:

- **Mild** An event is mild if the subject is aware of, but can easily tolerate the sign or symptom;
- **Moderate** An event is moderate if the sign or symptom results in discomfort significant enough to cause interference with the subject's usual activities;
- **Severe** An event is severe if the sign or symptom is incapacitating and results in the subject's inability to work or engage in their usual activities.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06

Page: 

#### 12.1.6 Device Deficiency

A Device Deficiency (DevD) is an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. DevD includes malfunctions, use errors and inadequate labelling.

#### 12.2 Reporting Procedures

AE of any kind and DevD will be recorded in the applicable CRF and source notes. The Investigator will evaluate all AE for relationship to the device and procedure, if applicable, seriousness, and severity. ADE, SAE, and DevD will be entered into the CRF and reported to the Sponsor within 24 hours of the investigator being informed about the event (Figure 12.2-1). For ADE and DevD, details of the product/procedure related to the event will be included and where applicable, pictures taken of the device. The deficient product should be retained for return to S&N unless it is contaminated (e.g. used dressings must not be retained). Updates to submitted information will be recorded in the CRF within 24 hours of the information being available to the investigator.

All SAE and ADE will be reviewed by a medically qualified person appointed by the Sponsor to determine which, if any, meet criteria for expedited reporting to the regulatory authorities.

The investigator will inform the IRB/IEC of adverse events according to the IRB/IEC requirements.

Depending on the nature of the adverse event, S&N may request copies of the subject's medical records, Imaging, Operative notes, as well as results of any relevant laboratory tests performed or other documentation related to the AE. If the subject was hospitalized, a copy of the discharge summary may be requested by S&N and should be forwarded as soon as it becomes available. In certain cases, S&N also may request a letter from the Investigator that summarizes the events related to the case. Refer to the ISF Sponsor Contact Information Sheet to report SAE, unanticipated ADE and SADE, anticipated SADE, and DevD.

# Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair | Smith&nephew | Number: 17-5010-06 | | Version: 1.0, 09/MAY/2018 | | Page: 

Figure 12.2-1: Evaluation and Reporting of AE and DevD



#### 12.3 Unblinding of Investigational Product

Not Applicable. This is an open-label study.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair > smith&nephew


Page: 

#### 12.4 FOLLOW-UP OF SUBJECTS WITH ADVERSE EVENTS

For subjects who are experiencing ongoing unresolved AE at the time of their study completion or early discontinuation from the study, it is recommended that the Investigator schedule an appropriate follow-up visit in order to determine the outcome of the event.

Any additional data must be documented and available to the Sponsor who will determine whether the data need to be documented within the CRF/Clinical Study Report.

#### 12.4.1 Ongoing Adverse Events at Study Discontinuation

Adverse events which are **related** to a study procedure or S&N IP and are ongoing at end of subject's participation: The event should be followed until it is either resolved or until the event has become chronic and is not expected to further improve based on Investigator's review of the event.

Adverse events which are **not related** to a study procedure or S&N IP and are ongoing at end of subject's participation should be followed for 30 days after discontinuation or if the AE is resolved, whichever is sooner.

At the time of data analysis (e.g. interim or final), an evaluation of ongoing events should take place and be listed as ongoing in the safety table.

#### 13. INVESTIGATOR OBLIGATIONS

The Principal Investigator (PI) will comply with the commitments outlined in the in the Statement of Investigator, provided by the Sponsor, and with Good Clinical Practice (GCP), and all applicable regulatory requirements as outlined in Appendix 21.4 of this protocol.

In addition, the PI will ensure that the Financial Disclosure Statements will be completed by the PI and the Sub-Investigator upon entry into the study and as any changes that affect their

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair smith&nephew


Page: 

financial disclosure status occur during the course of the study and up to one year after study completion.

#### 14. SPONSOR AND MONITOR RESPONSIBILITIES

The Sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals. The clinical investigation will be monitored to ensure that: the rights and wellbeing of the subjects are protected; the reported data are accurate, complete, and verifiable from the source documents; and the study is conducted in compliance with the currently approved protocol, with GCP regulations, and with applicable regulatory requirements.

Detailed monitoring requirements will be documented within the Clinical Monitoring Plan for this study.

#### 14.1 CONTRACT RESEARCH ORGANIZATION

The Sponsor has engaged Contract Research Organization (CRO) to assist in conducting this study. When appropriate, the CRO is referred in study documents as "Sponsor's agent".

#### 14.2 SITE QUALIFICATION VISIT

A site qualification visit may be performed by the Sponsor prior to the execution of a clinical agreement to ensure that all Investigators have the appropriate training, staff, facilities, and resources to adequately conduct the study.

#### 14.3 SITE INITIATION VISIT

A site initiation visit to provide training on the specifics of the study, site obligations and expectations of study conduct will be performed by the Sponsor or qualified person designated by the Sponsor following the execution of the CTA (Clinical Trial Agreement) and documented IRB/IEC approval.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair smith&nephew


**Page:** 

#### 14.4 Sponsor Audits and Regulatory Inspection

Quality Assurance auditors, whether an employee of the Sponsor or its designee, may evaluate study conduct at the study sites. These parties must have access to any and all study reports and source documentation, regardless of location and format.

#### 14.5 CLOSE-OUT VISIT

A study close-out visit will be performed by the Sponsor or designee to retrieve and account for all remaining clinical data and to resolve outstanding queries. During study close-out, the monitor will review investigator files to ensure required documents and records are on file, and review regulatory requirements regarding records retention and IRB/IEC reporting requirements.

#### 15. PROTOCOL AMENDMENTS

Amendments should be made only in exceptional cases once the study has started. Protocol amendments must be approved by the protocol signatories prior to submission to the IRB/IEC. Protocol amendments need to be approved by the IRB/IEC and Regulatory Authority(ies), as applicable prior to implementation at the site

#### 16. CONFIDENTIALITY OF THE STUDY

The confidentiality of this study and associated documents is governed by the terms of the Clinical Trial Agreement (CTA).

#### 17. STATEMENTS OF COMPLIANCE

This clinical study will be performed in compliance with the ethical principles of the Declaration of Helsinki; ISO 14155:2011 Clinical investigation of medical devices – Good Clinical Practice; ICH-E6.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

This clinical study will not commence until the required approval/favorable opinion from the IRB/IEC or regulatory authority has been obtained. Any additional requirements imposed by the IRB/IEC or regulatory authority will be followed.

Public/Products Liability Insurance has been purchased by Smith & Nephew plc. Worldwide and incorporates coverage for personal injury in respect of clinical studies. The Sponsor agrees to operate in good faith and in accordance with ABHI (Association of British Healthcare Industries) guidelines regarding compensation for injury arising in the course of clinical studies.

#### 18. END OF STUDY

The end of the study is defined by the last visit of the last subject undergoing treatment in the study.

#### 19. PUBLICATION POLICY

#### 19.1 Publication of Study Data

The preparation and submission for publication of manuscripts containing the study results shall be in accordance with a process determined by the Clinical Trial Agreements between the study Sponsor and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws, including, but not limited to the Health Insurance Portability and Accountability Act of 1996.

#### 19.2 DATA SHARING

Smith & Nephew is committed to upholding the highest ethical and legal standards involved in conducting clinical trials. Smith & Nephew therefore supports the data sharing requirements of The International Committee of Medical Journal Editors (ICMJE) published on the 6th June 2017. In accordance, Smith & Nephew will consider requests to share individual (deidentified) participant data that underlie the results of any interventional clinical trial, as presented from the 1st July 2018 within an ICMJE associated journal. Requests made by researchers who provide a

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Page:** 

methodologically sound proposal will be considered. Requests may include data that underlie results presented in text, tables, figures and appendices, together with data dictionaries. Availability of these data will begin 9 months and end 36 months after article publication. Data supplied may only be used by the researcher(s) named in the approved research proposal for the purposes of achieving the aims of the analyses specified therein. All proposals should be directed to <a href="mailto:datasharing.gcs@smith-nephew.com">datasharing.gcs@smith-nephew.com</a>. To gain access, data requestors will need to sign a data access agreement.

#### 20. REFERENCES

- Demehri S, Hafezi-Nejad N, Fishman EK. Advanced imaging of glenohumeral instability: the role of MRI and MDCT in providing what clinicians need to know. *Emergency radiology*. 2017;24(1):95-103.
- Erickson J, Lavery K, Monica J, Gatt C, Dhawan A. Surgical treatment of symptomatic superior labrum anterior-posterior tears in patients older than 40 years: a systematic review. Am J Sports Med. 2015;43(5):1274-1282.
- 3. **Werner BC, Brockmeier SF, Miller MD**. Etiology, Diagnosis, and Management of Failed SLAP Repair. *The Journal of the American Academy of Orthopaedic Surgeons*. 2014;22(9):554-565.
- 4. **McCormick F, Bhatia S, Chalmers P, Gupta A, Verma N, Romeo AA**. The management of type II superior labral anterior to posterior injuries. *The Orthopedic clinics of North America*. 2014;45(1):121-128.
- 5. **Zlatkin MB, Sanders TG**. Magnetic resonance imaging of the glenoid labrum. *Radiologic clinics of North America*. 2013;51(2):279-297.
- 6. **Rossy W, Sanchez G, Sanchez A, Provencher MT**. Superior Labral Anterior-Posterior (SLAP) Tears in the Military. *Sports health*. 2016;8(6):503-506.
- 7. **Tayrose GA, Karas SG, Bosco J**. Biceps Tenodesis for Type II SLAP Tears. *Bulletin of the Hospital for Joint Disease (2013)*. 2015;73(2):116-121.
- 8. **Griffin JW, Leroux TS, Romeo AA**. Management of Proximal Biceps Pathology in Overhead Athletes: What Is the Role of Biceps Tenodesis? *American journal of orthopedics (Belle Mead, N.J.).* 2017;46(1):E71-e78.
- 9. **Vianello R, Pannone A, Conca M, Corezzola R**. Return to Sport After Shoulder Arthroscopy. In: Volpi P, ed. *Arthroscopy and Sport Injuries: Applications in High-level Athletes*. Cham: Springer International Publishing: 2016:175-184.
- 10. **Smith MV, Calfee RP, Baumgarten KM, Brophy RH, Wright RW**. Upper Extremity-Specific Measures of Disability and Outcomes in Orthopaedic Surgery. *The Journal of Bone and Joint Surgery. American volume*. 2012;94(3):277-285.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06
Page: 

- 11. **Mook WR, Briggs KK, Philippon MJ**. Evidence and Approach for Management of Labral Deficiency: The Role for Labral Reconstruction. *Sports medicine and arthroscopy review.* 2015;23(4):205-212.
- 12. **Ayeni OR, Adamich J, Farrokhyar F, et al.** Surgical management of labral tears during femoroacetabular impingement surgery: a systematic review. *Knee surgery, sports traumatology, arthroscopy: official journal of the ESSKA.* 2014;22(4):756-762.
- 13. **Fayad TE, Khan MA, Haddad FS**. Femoroacetabular impingement: an arthroscopic solution. *The bone & joint journal*. 2013;95-b(11 Suppl A):26-30.
- 14. **Kollmorgen R, Mather R**. Current Concepts in Labral Repair and Refixation: Anatomical Approach to Labral Management. *American journal of orthopedics (Belle Mead, N.J.).* 2017;46(1):42-48.
- 15. **Skendzel JG, Philippon MJ**. Management of labral tears of the hip in young patients. *The Orthopedic clinics of North America*. 2013;44(4):477-487.
- 16. **Wolff AB, Grossman J**. Management of the Acetabular Labrum. *Clinics in sports medicine*. 2016;35(3):345-360.
- 17. **El Bitar YF, Lindner D, Jackson TJ, Domb BG**. Joint-preserving surgical options for management of chondral injuries of the hip. *The Journal of the American Academy of Orthopaedic Surgeons*. 2014;22(1):46-56.
- 18. **Khan M, Bedi A, Fu F, Karlsson J, Ayeni OR, Bhandari M**. New perspectives on femoroacetabular impingement syndrome. *Nature reviews. Rheumatology.* 2016;12(5):303-310.
- 19. **Salata MJ, Vasileff WK**. Management of Labral and Chondral Disease in Hip Preservation Surgery. *Sports medicine and arthroscopy review.* 2015;23(4):200-204.
- 20. **Kivlan BR, Nho SJ, Christoforetti JJ, et al.** Multicenter Outcomes After Hip Arthroscopy: Epidemiology (MASH Study Group). What Are We Seeing in the Office, and Who Are We Choosing to Treat? *American journal of orthopedics (Belle Mead, N.J.).* 2017;46(1):35-41.
- 21. **Agrawal V, Pietrzak WS**. Triple labrum tears25. repaired with the JuggerKnot soft anchor: Technique and results. *Int J Shoulder Surg.* 2015;9(3):81-89.
- 22. **Boileau P, Gendre P, Baba M, et al.** A guided surgical approach and novel fixation method for arthroscopic Latarjet. *Journal of Shoulder and Elbow Surgery.* 2015.
- 23. **Matsuda DK, Gupta N, Burchette RJ, Sehgal B**. Arthroscopic surgery for global versus focal pincer femoroacetabular impingement: are the outcomes different? *Journal of Hip Preservation Surgery*. 2015:hnv010.
- 24. **Agrawall V, Pietrzak WS.** Triple labrum tears repaire with the JunggerKnot soft anchor: T Technique and results. *Int J Shoulder Surg.* Jul-Sep 2015;9(3):81-89
- 25. **Peacock JL, Kerry S.** Presenting medical statistics from proposal to publication: a step-by-step guide. Oxford University Press; 2007.
- 26. **Lafosse, L., Brzoska, R., Toussaint, B. and Gobezie, R., 2008.** The outcome and structural integrity of arthroscopic rotator cuff repair with use of the double-row suture anchor technique. *J Bone Joint Surg Am*, (Supplement 2 Part 2), pp.275-286.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair \*\*Smith&nephew
Number: 17-5010-06

**Page:** 

- 27. **Salaffi F, Sarzi-Puttini P, Atzeni F. Best Pract Res Clin Rheumatol.** 2015 Feb;29(1):164-86. doi: 10.1016/j.berh.2015.04.023. Epub 2015 Jun 19. Review.
- 28. ISO 14155:2011
- 29 CFR 812
- 30. ICH Guideline for Clinical Safety Data Management: Definitions and Standards for Expedited Reporting

| Study Protocol—Device | smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market Clinical Follow-<br>up Study to evaluate safety and performance of the | Number: 17-5010-06<br>Version: 1.0, 09/MAY/2018 |
| SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair | Page: |

## 21. APPENDICES

21.1 INSTRUCTIONS FOR USE SUTUREFIX ULTRA AND SUTUREFIX CURVED

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06


Page: 

#### > smith&nephew

SUTUREFIX Ultra Suture Anchor



EG REP Hull HUS SSN United Kingdom ocrop@amith-nog



(€...

00/0017 10401050 Per D

#### SUTUREFIX Ultra Suture Anchor

SUTURERX Ultra Fadenanker

Anclaie para suturas SUTURERX Ultra Ancrage de suture SUTURERX Ultra Ancora di sutura SUTURERX Ultra SUTURERX Ultra suturankare SUTURERX Ultra hechtdraadanker Ancora de sutura SUTURERX Ultra SUTURERX Ultra suturanker SUTURERX Ultra suturanker SUTURERX Ultra 봉합사고정기

Instructions for Use Mode d'emplo istruzioni per l'uso Bruksanvisning Gebruksaanwijzing instruções de utilização Brugsanvisning Bruksanvisning 사용 지설

English

#### SUTUREFIX Ultra Suture Anchor

② STERILE EO 

■

#### Device Description

Desvice Dessil priorii

The Smith & Niephow SUTUSKX (thre Suure ûnchor is
a floation douter intended to provide accuration to
affit thas to brone. It consists of a affit actus annoter
with attached non-standard actually pressure fisch
an inscrite not obtain. The anchors are antialistic provided
with other one of autore or two fill subtree. This debtails
provided sending, for antiglic uses of the
provided sending, for antiglic uses one.

#### Contents

- Non-absorbablo suturo anchor-bratdod, afloono exated, pdyrater (USP), non-absorbablo

Braidad, uncostod,UHWWpolydhylana, white and/or blue, non-absorbable and/or

UHWW golydhylana with manofilamentnylan cobraid (black), nan-absobable

Refer to Individual auture anchor greduct labels for autus size, type, and quantities.

#### Indications for Use

Hip capaulo repair

#### Shoulder

- Bankert ropatr
- Antorior shouldor instability SAP loston regains
- Cansular shift or cansulolabral reconstructions
- Dohold regains
- Bloops tonodosts

#### Foot and Ankle

- Hallus valgus regate
- Model or lateral tratability regards
- Achillos tandan regal/s/reconstructions Midfoot reconstructions
- Motatarsal ligamort/tandon regalita/reconstructions

#### Elbow, Wrist, and Hand

- . Unar or radal colatoral ligament reconstructions Latoral optoordylitis ropat

- Model coletoral ligament
   Lateral coletoral ligament
- Postorior obliguo ligament
- Patolar roslignmentand tenden regalns
   Vastus modells obliguus advancement
- Notibial band tonodosis

#### Contraindications

- Known hygoracosithity to the implant material. Who material sensithity is auspected, appropriate tests should be performed and sensitively suice outprior to implantation.
- Pathological conditions of bono, such as oatic changes or source esteepers, which would compromise secure anchor floation.

19601039. Ror R

#### A Warnings

- Contents are sterile unless package to opened or damaged, DO NOT RESTERUES, For single use only. Discard any open, unused product. Oc-use, after the expiration date.
- It is the surgeon's exponsibility to be familiar with the appropriate surgical techniques prior to use of this device.
- Read these instructions completely prior to use.
- Maintaining guide alignment throughout drilling to required to ensure drill bit integrity.
- Do not reaterfize or reuse anchors, suturesed insertion devices packaged with the anchor.
- incomplete anchor insertion may result in por anchor performance.

#### Precautions

P<sub>A</sub> U.S. Fodoral law catricts this dovice to sale by even on the order of aphysician.

- Hazards seasolated with rouse of this de-tecinolude, but are not limited to gattent infaction and/or device marginetics.
- Prior to use, inspect the device to ensure it is not demaged. Do not use a damaged device.
- Postoporative case is important, instructife gallet on the limitations of the implant and saution from regarding weight bearing and body stresses onto appliance grier to secure bone healing.
- Do not uso sharp instruments to manage or control the suture.
- to source.

  As with any source anchor or sourcing technique, the floation given whold be considered as only temperary, will biological attachment for insue to bone to completed, and may not eitherstend using bearing or other unapported streams. The salue anchor and source are not insued to ground indepints biomochantal integrity.
- Implantation of the sature archerogules proparation of the insertion site Prodelling with the appropriate Smith & Nephew Drill Sit is the preferred method of site proparation.
- Ensure the archer placement is aligned with the drilled hole. Proper alignment is easential for successful repair.
- Use of excessive force during insertion can cause failure of the suture anchor or insertion device.
- Bono quality must boardoquate to allowgrops placement of the autorearcher.

- Postogorative range of motion is to be determined by the physician.
- After use, this dovice may be a getential blokscard and should be handled in accordance with accepted medical gractice and applicable local and national regulerements.

#### Adverse Reactions

- Mid inflammatory reaction
- Foreign body reaction
- nfaction, both doop and suporficial
- Alloreto rosistion

#### Instructions for Use

Note: Use the appropriate Smith & Nephow Instrumentation is necessary to proper the insertion ato and maintain sotal alignment between the insertion also and the SUTURERY Utra Subrealador.

- Soloct the appropriate auture anchor instrument length (S or XI), based on the apositic indication proformed surgical technique, and patient history

Hold the drill guide firmly in place and use the appropriate auture anchor drill bit to propare the transition site. The depth step on the drill bit betters out on the handle of the drill guide when proper table doubt is reached.

| Dull Gride | DHI BR | Anchor |
|------------|-----------|-----------|
| S | 1.7 mm S | 1.7 mm S |
| XL | 1.7 mm XL | 1.7 mm XL |
| 5 | 1.0 mm S | 1.0 mm S |

- Instrumentation is available in the longfix standard (S) and extralong XIL. Sdootfie drift that corresponds with the guide. Hold the drift guide stack, maintain alignment, and remove the drift list from the insection site. Verify that the drift list is notating forward.
- the one of a reason covers.

  Continue to had the dill guide firmly in place and insent the auture anchor into the guide with the dealted auture orientation. To insent the anchor:
- positions the auture anchor to the appropriate dopth below the surface of the bone.

CAUTION: Do not rotate the auture anchordentee once seated in the bone as this may cause deter

Koop the drill guide in place and grow the lack button on the handle to unlock the sliding ring





Aguve, As., Suturcendror Agure 16. Suturcendror hendio (pro-doployment) hendio (post-doployment)

- Doploy the anchor by pulling back on the alding ring until a clickle hand. This click confirms proper anchor diployment Figure 1b;
- Unwind the suture from the new exposed suture cleat.
- waterion dovice from the distinguide. The andre will remain in the bone and the auture will feet through the handle as it is removed.
- a. Discard the insertendevia:
- CAUTION: After use, this delice maybe a potential biohazard and should be hardled in accordance with acsigner medical gradicea applicable local and national requirements.

- or the auture and/or in the implantation site.

  Pass the registratures frought arrest middle status to be reflected uning the desired auture gassing to configure and desires.

  Secure the regain of the fissue with standard lend tying techniques without members, cut and immost any occess auture.
- 10 Place additional auture anchors as regulad to complete the procedure.

#### Warranty

For Further Information

if further information on this product is needed, contact Smith & Nephow Customer Senice at 41,800,848,550 In the U.S., or an authorized representative.

#4004.60039nthAlaphy.log Alingtonomed

10401059 Rev 9

10401049.764

SUTURGEX Ultre Sauro.indro Instructions for Us

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06


**Page:** 

#### smith&nephew

SUTUREFIX® Curved Suture Anchor



EC REP EuropeanRepresentative Smith & Nophow Hodical United 101 Hopes, Road Hus HUS SEN





SUTUREFIX® Curved Suture Anchor

SUTURERX gebogenerFadenanker Anclaje curvado para suturas

Ancrage de suture incurvé SUTURERX Ancora di sutura curva SUTURERX SUTURERX Böit suturankare

SUTURERX gebogen hechtdraadanker Ancora de sutura curva SUTURERX SUTURERX Buetsuturanker

SUTURERX buet suturanker SUTURERX 곡선형 봉합사고정기

Изогнутый шовный якорь SUTURERX

SUTUREFIX Kıvrık Sütür Kancası

#### Instructions for Use Gebrauchsanweisung

Modo de empleo Mode d'emploi Istruzioni per l'uso Bruksanvisning Gebruiksaanwijzing Instruções de utilização

Bruksanvisning 사홉 지설

Инструкция поприменению Kullanım Talimatları



Illiangrote rezeranci sub + III.-goolgrot
III.grotevanend + Seguro paragrocedinistració
Sil incorrenta magnifica i Continue sucrimorea de
diautifica na independia i III. della magnificante con adultation de la continue del la continue de la continue del la continue de la cont

English

SUTUREFIX® Curved Suture Anchor



#### Contents

Non-ebsorbeblo suluro endror - breidzij alicono certod poljostor IUSPI, gopostastiskabilo,

CarGos: Subres-Breided, uncoaled, UHIIN poljetylene, white

Rofor to includual suluro anchor productlabolator suluro ato, tipo, and quantitios.

#### Intended Use

#### Indications for Use

The Smith & NephewSUTURENC Curried Subtrackathers are intended for the assure faster of soft faste observe for the following indications.

#### Shoulder Cognition stabilization

- Sentertropeir
- Anterior shoulder instability SLAP loaten regelra.

#### Contraindications

- When ingranding to be ingleninaterial. Who matrial smalling is supported, appropriate total about the performance and smallingrude outgrothe inglenation.

  Pathological conditions of bone, such as signific divergence reserve categories, which incuid compromise source categories, which incuid compromise source and or faster.
- Pethological conditions in the soft fissues to be attached that heald impet accurs factor by subre. Comminuted bone surisce, which would compromise source anchor factor.

#### A Warnings

Do not use if padage is damaged. Do not use if the product sterification barrier or hapadaging is compromised.

- Contentrare sterile unless gadage is opened or damaged, DO NOT RESTRUCE. For single use only. Discard anyopen, unused product. De, menuse, after the expiration date.
- after the expiration date.

  Prior to use, inspect the product padage for crucional integrity. If the east of the outer diefe barrier is broken, or if the death barrier tearns otherwise damaged, the product should be conditioned non-marks and not be used.
- It is the surgeon's regionability to be times re-the appropriate anglish rediniquesprish to use this deate. Read these instructions completely prior to use. Productinus be stored in the original easied pouts. Incomplete ander heartion may result in the ander not functioning as intended.

- Greatings of the faible Interter can occur if the interter can occur if the intertion do is not prepared with recommended smith & Haphew curried guide & faible criti prior to hearties.

SUTURISTIC Curried Suture Anchor Instructions for Use

English

- Haintaining guide alignment throughout drilling is required to ensure drill bit integrity. Do not attempt to implant this deales within cartiage epiphysisal growth planeaut non-ceasous tissue.

#### Precautions

- $\underline{\underline{R}}_{i}$  U.S. Redoral law restricts this device to said by error the order of a physician.
- a make and projected.

  Heards excelleted with rouse of his device include, but are not limited to geten this clien and/order mellunden.
- metunation.

  Prior to use, inspect the device to ensure trained demagnd. De not use a demagnd device.

  Postoperatio sare talegoriant instruct the patient on the limitations of the implantand surfain from regarding veightboaring and body stresses on the appliance prior to secure bone healing
- the suture. Is with any suture enther or suturing technique, the feation given should be considered as only temperary, unfill-bloogical attechment of feation to bone is completed, and may not with attend weight. boaring or other unsupported stresses. The sulue endher and sulure are not intended to greated indefinite blomechanical integrity.
- Indefine blemederical integrity, implementation than always earth agreement of the active author requires green of the facilities with the aggreement of the facilities of the
- Use of executive force during insertion cancause failure of the suture enchor or insertion device.
- Sono quality must be adequate to allow grops placement of the auture anchor.
- giscomentation subtrainments of phonoisments of the contract of the inglander information performance maybe admensional performance maybe admensionable.

  Once see the discontract to the subtrainments of the contract of the
- Wor use, this device may be a potentialblohasard and should be handled in accordance with accepted modical gradice and applicable local and national requirements.

#### Adverse Reactions

- Loss officetion or cultout of suturo encharace noccur IIIId infermetoryroadon

#### Instructions for Use

Note: Use the appropriate Smith & Neghow Instrumentation is necessary to propere the insertion ate and maintain satal alignment between the insertion ate and the SUTURSPY, Curried Suturalization.

Note: The following SUTURSEX: Curried instruments and

| Drill Guide | DVE SH | Anthor |
|-------------|----------|----------|
| s | 17mm S | 17 mm S |
| XL. | 17mm XL | 17mm XL |
| S | 1.9 mm S | 1.9 mm S |

instrumentation is evaluable in the longths standard SI and extra-long 00. Select the drill the corresponds with

- Place the district ty of the curred drill guide onto the bone eithe desired implantation site. Curred Drill guide placement may be alded using an optional fecible obtunator.

Note: For dones bono, timey bo required togido the featble, drill in and out of the implantation afte to

1060%58 Rev&

English

- Hold the curred drill guide abody, maintain alignment and remove the featble drill bit from the insertion afte. CAUTION Conclumers the cursed distinguide from the onder inaction site.
- Continue to hold the curred drill guide firmly in place and inserting facilities suffer and/or into the curred guide with the deathed suffer prioritation. To insertite anchon.
- Note: If tagging, uso multiple light tagging controlled insertion.
- continue to guide or tog until the anchor handle makes contact with the curred drill guide handle. This positions the subre anchor to the appropriate depth below the surface of the bone.

CAUTION Do not rotes the auture onder distar once social in the boness this may course distar follow. Doploy the suburo anchor.

Koop to curred drill guide in place and prossitio lock buffer on the handle to unlock the stiding ring Reuro Isl.





Rouge to Surtreandorhardispost-dag

c. Unwind the suture from the newexposed suture doet.

o. Dispard the insertion device.

c. Dissert the insert notice.
CAUTION: After use, the deter maybe a potential blothcost and stoud to thended in coordance with coupled maintain produce and applicable local and notional equitments.
Rougely brains to the subure to confirm the stability of the subure endors in the subure to sometime the subure of the subure and/or in the legislands on the.

- Pess the regain subtreathrough or around the set tasks to be established using the desired subtrepessing
- Secure the regain of the faster with standard lines tying techniques. When complete, cut andrenese

Warranty

For Further Information If further information on this groduct is needed, contact Smith & Nephow Customer Sonito at 41, 800, 949, 277 In the U.S., or an authorized regressivative.

Tradomatic/Shift & Nighow, egisteedU.S. Patent& TradomaticNto. 96017 Shift & Nighov, Inc. All fighterapence.

SUTURISTIC Curried Sulture Anchor Instructions for Use 10601656868

| Study Protocol—Device | smith&nephew |
|---|---|
| Prospective, Multicenter, Post-Market Clinical Follow- | Number: 17-5010-06 |
| up Study to evaluate safety and performance of the | <b>Version:</b> 1.0, 09/MAY/2018 |
| SUTUREFIX ULTRA and SUTUREFIX CURVED Suture | Page: |
| Anchors in shoulder and hip arthroscopic repair | |

### 21.2 PROTOCOL AMENDMENT

Not applicable, this protocol has not been amended.

# Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair | Smith&nephew | Number: 17-5010-06 | | Version: 1.0, 09/MAY/2018 | | Page: 

#### 21.3 QUALITY OF LIFE MEASURES EQ-5D-5L

Under each heading, please tick the ONE box that best describes your health TODAY.

| MOBILITY |
|---|
| I have no problems in walking about |
| I have slight problems in walking about |
| I have moderate problems in walking about |
| I have severe problems in walking about |
| I am unable to walk about |
| SELF-CARE |
| I have no problems washing or dressing myself I have slight problems washing or dressing myself |
| I have moderate problems washing or dressing myself |
| I have severe problems washing or dressing myself |
| I am unable to wash or dress myself |
| USUAL ACTIVITIES (e.g. work, study, housework, family or |
| leisure activities) |
| I have no problems doing my usual activities |
| I have slight problems doing my usual activities |
| I have moderate problems doing my usual activities |
| I have severe problems doing my usual activities |
| I am unable to do my usual activities |
| PAIN / DISCOMFORT |
| I have no pain or discomfort |
| I have slight pain or discomfort |
| I have moderate pain or discomfort |
| I have severe pain or discomfort |
| I have extreme pain or discomfort |
| ANXIETY / DEPRESSION |
| I am not anxious or depressed |
| I am slightly anxious or depressed |
| I am moderately anxious or depressed |
| I am severely anxious or depressed |
| I am extremely anxious or depressed |

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair smith&nephew

Number: 17-5010-06


Page: 

- . We would like to know how good or bad your health is TODAY.
- . This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- . Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =



Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06


Page: 

#### 21.4 ADDITIONAL ASSESSMENTS

#### **Patient Hip Assessments**

#### Pain Assessment

1. Please select a number from the scale below that indicates the level of pain you are experiencing from your hiptoday



\*Please provide a reason for your score \_

#### Patient Satisfaction

2. Please select a number from the scale below that indicates your level of satisfaction with the arthroscopy repair surgery to stabilize your <u>hip</u>



\*Please provide a reason for your score

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06


**Page:** 

#### Patient Shoulder Assessments

#### Pain Assessment

1. Please select a number from the scale below that indicates the level of pain you are experiencing from your shoulder today



\*Please provide a reason for your score \_

#### Patient Satisfaction

2. Please select a number from the scale below that indicates your level of satisfaction with the arthroscopy repair surgery to stabilize your <u>shoulder</u>



\*Please provide a reason for your score \_

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

| > smitn&nepnew |
|--------------------------|
| Number: 17-5010-06 |
| Version: 1.0.00/MAY/2018 |

Page: 

1

Hip dysfunction and Osteoarthritis Outcome Score (HOOS), English version LK 2.0

| the dystalicidal and Ostobalianitis Outcome Score (11000); English Velsion Enc. 20 | | | | |
|---|---|---|---|---|
| HOOS HIP SURVEY | | | | |
| | | | | _ |
| Today's date: | !! | Date of birth: | | |
| Name: | | | | |
| will help us keep t<br>your usual activitio | track of how you<br>es.<br>estion by ticking t | feel about your h<br>the appropriate b | ip and how well y<br>ox, only <u>one</u> box | for each question. |
| Symptoms<br>These questions s<br>during the last we | | ered thinking of y | our hip sympton | ns and difficulties |
| S1. Do you feel grin | ding hear clicking | g or any other type o | of noise from your l | nip? |
| Never | Rarely | Sometimes | Often | Always |
| S2. Difficulties spre | ading legs wide ap | art<br>Moderate | Severe | Extreme |
| S3. Difficulties to st | | | | <b>.</b> |
| None | Mild | Moderate | Severe | Extreme |
| 0 | | | | <u> </u> |
| Stiffness The following que during the last we the ease with which | <b>ek</b> in your hip. St | tiffness is a sensa | | |
| S4. How severe is y | our hip joint stiffn | ess after first waker | ning in the morning | ? |
| None | Mild | Moderate | Severe | Extreme |
| S5. How severe is y | our hip stiffness af<br>Mild | fter sitting, lying or: | resting later in the<br>Severe | day? |
| _ | _ | _ | _ | _ |
| Pain | | | | |
| P1. How often is you | | | | |
| Never | Monthly | Weekly | Daily | Always |
| □<br>What amount of hactivities? | nip pain have yo | ou experienced th | ne last week dur | ing the following |
| P2. Straightening yo | our hip fully | | | |
| None None | Mild | Moderate | Severe | Extreme |

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

Number: 17-5010-06

**Version:** 1.0, 09/MAY/2018 Page: 

| Hip dysfunction and Osteoarthritis Outcome Score (HOOS), English version LK 2.0 | | | | |
|---|---|---|---|---|
| What amount of hip activities? | pain have yo | ou experienced th | ie <b>last week</b> dui | ring the following |
| P3. Bending your hip f | ully | | | |
| None | Mild | Moderate | Severe | Extreme |
| P4. Walking on a flat s | urface | | | |
| None None | Mild | Moderate | Severe | Extreme |
| P5. Going up or down | stairs | | | |
| None | Mild | Moderate | Severe | Extreme |
| | | | _ | |
| P6. At night while in b | | | | |
| None | Mild | Moderate | Severe | Extreme |
| | | 0 | | |
| P7. Sitting or lying | | | | |
| None | Mild | Moderate | Severe | Extreme |
| P8. Standing upright | | | | |
| None | Mild | Moderate | Severe | Extreme |
| P9. Walking on a hard | surface (asphalt | concrete etc.) | | |
| None | Mild | Moderate | Severe | Extreme |
| | | | _ | |
| P10. Walking on an un | | | | |
| None | Mild | Moderate | Severe | Extreme |
| Function, daily living The following questions concern your physical function. By this we mean your ability to move around and to look after yourself. For each of the following activities please indicate the degree of difficulty you have experienced in the last week due to your hip. | | | | |
| A1. Descending stairs | | | | _ |
| None | Mild | Moderate | Severe | Extreme |
| A2. Ascending stairs | | | | |
| None | Mild | Moderate | Severe | Extreme |
| A3. Rising from sitting | | | | |
| None | Mild | Moderate | Severe | Extreme |
| A4. Standing | | | | |
| None | Mild | Moderate | Severe | Extreme |
Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

| > smith&nephew |
|----------------|
|----------------|

**Number:** 17-5010-06

3

**Version:** 1.0, 09/MAY/2018 **Page:** 

Hip dysfunction and Osteoarthritis Outcome Score (HOOS), English version LK 2.0

For each of the following activities please indicate the degree of difficulty you have experienced in the **last week** due to your hip.

| A5. Bending to the | floor/pick up an o | bject | | |
|---|---|---|---|---|
| None | Mild | Moderate | Severe | Extreme |
| | | 0 | | |
| A6. Walking on a f | lat surface | | | |
| None | Mild | Moderate | Severe | Extreme |
| 0 | | | | |
| A7. Getting in/out | of car | | | |
| None | Mild | Moderate | Severe | Extreme |
| A8. Going shoppin | g | | | |
| None | Mild | Moderate | Severe | Extreme |
| | | | 0 | |
| A9. Putting on sock | ks/stockings | | | |
| None | Mild | Moderate | Severe | Extreme |
| 0 | | | | |
| A10. Rising from b | | | _ | _ |
| None | Mild | Moderate | Severe | Extreme |
| A11. Taking off so | | | | _ |
| None | Mild | Moderate | Severe | Extreme |
| A12. Lying in bed ( | (turning over, mai | ntaining hip position) | ) | |
| None | Mild | Moderate | Severe | Extreme |
| A13. Getting in/out | of bath | | | |
| None | Mild | Moderate | Severe | Extreme |
| | | | 0 | |
| A14. Sitting | | | | |
| None | Mild | Moderate | Severe | Extreme |
| 0 | | | | |
| A15. Getting on/off | | | | <b>.</b> |
| None | Mild | Moderate | Severe | Extreme |
| | | heavy boxes, scrubb | | |
| None | Mild | Moderate | Severe | Extreme |
| A17. Light domesti | | | Conse | Posteron |
| None | Mild | Moderate | Severe | Extreme |

during the last week due to your hip.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

| > smith&nephew |
|---------------------------|
| Number: 17-5010-06 |

**Page:** 

4

| | | _ | | | |
|---|---|---|---|---|---|
| Hip dysfunction | and Osteoarthritis | s Outcome Score | (HOOS). | English vers | ion LK 2.0 |

Function, sports and recreational activities
The following questions concern your physical function when being active on a higher level.
The questions should be answered thinking of what degree of difficulty you have experienced

| SP1. Squatting<br>None | Mild | Moderate | Severe | Extreme |
|---|---|---|---|---|
| SP2. Running | | | | |
| None | Mild | Moderate | Severe | Extreme |
| SP3. Twisting/pivot | ing on loaded leg | | | |
| None | Mild | Moderate | Severe | Extreme |
| SP4. Walking on un | even surface | | | |
| None | Mild | Moderate | Severe | Extreme |
| Quality of Life | | | | |
| Q1. How often are y | ou aware of you | rhip problem? | | |
| Never | Monthly | Weekly | Daily | Constantly |
| Q2. Have you modif | fied your life styl | e to avoid activities p | otentially damagin | g to your hip? |
| Not at all | Mildly | Moderately | Severely | Totally |
| | ٥ | | | |
| Q3. How much are y | you troubled with | lack of confidence in | ı your hip? | |
| Not at all | Mildly | Moderately | Severely | Extremely |
| Q4. In general, how | much difficulty | do you have with you | r hip? | |
| None | Mild | Moderate | Severe | Extreme |

Thank you very much for completing all the questions in this questionnaire.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06


Page: 

#### Modified Harris Hip Score (mHHS) Calculation SOURCE WORKSHEET

| Clinician Name: |
|---------------------|
| Subject ID: |
| Subject Code: |
| Date (DD/MMM/YYYY): |

#### Instructions:

Use this Work Instruction as source documentation for the total mHHS calculation (mHHS question 12). The total mHHS is considered NULL if any question 1-8 is missing. mHHS questions 9-11 are not included in the total mHHS calculation.

Enter the actual score for questions 1-8 that correlates to the study subject's mHHS questionnaire response. To obtain the total mHHS add the actual scores from questions 1-8 then multiply by 1.1.

| | Possible | Actual |
|----------------------------------------------|----------|--------|
| Question | Score | Score |
| 1. Hip Pain: | | |
| none or ignores it | 44 | |
| slight, minimal; no compromise in activities | 40 | |
| mild; following longer activities | 30 | |
| moderate; some limitations of activities | 20 | |
| marked; serious limitations of activities | 10 | |
| Disabled; no activities possible, bedridden | 0 | |
| 2. Enter public transportation: | | |
| yes, possible | 1 | |
| no, unable | 0 | |
| 3. Putting on shoes and socks: | | |
| with ease | 4 | |
| with difficulty | 2 | |
| unable | 0 | |
| 4. Distance walked: | | |
| unlimited, several hours | 11 | |
| six blocks, up to 2 km/1 mile | 8 | |
| daily shopping, up to 500 km/.3 miles | 5 | |
| indoors only, up to 50 m/150 feet | 2 | |
| bed / chair / not able to walk | 0 | |

| | Possible | Actual |
|---------------------------------------------|----------|--------|
| Question | Score | Score |
| 5. Support: | | |
| None | 11 | |
| single cane for long walk | 7 | |
| single cane most of the time | 5 | |
| one crutch | 3 | |
| two canes | 2 | |
| two crutches or not able to walk | 0 | |
| 6. Stairs: | | |
| foot over foot, without banister | 4 | |
| foot over foot, with banister | 2 | |
| in a manner | 1 | |
| unable | 0 | |
| 7. Sitting: | | |
| comfortably in any chair for one hour | 5 | |
| comfortably on high chair for one-half hour | 3 | |
| unable to sit comfortably | 0 | |
| 8. Limp: | | |
| none | 11 | |
| slight | 8 | ] |
| moderate | 5 | |
| severe | 0 | |
| Questions 1-8 Total: | | |
| Total mHHS (Questions 1-8 Total x 1.1): | | |

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 



Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

| >!- | smith | &nei | hew |
|-----|----------|------|-------|
| 1 | SIIIIIII | απε | JIIEW |

Number: 17-5010-06 Version: 1.0, 09/MAY/2018 Page: 

| > smith&nephew <study pg="" title@master=""> XX-XXXX-XX</study> | Constant Shoulder Score<br>(CSS) | Subject ID: Left Right |
|---|---|---|
| INSTRUCTIONS: Please select of During the past 4 weeks | ne answer from each of the following qu | estions. |
| 1. Pain Severe Moderate Mild None 3. Arm positioning Up to waist Up to xiphoid Up to neck Up to top of head Above head | Full re Full w 4. Stren 0 1- 4- 7- | Yes No ected sleep |
| RANGE OF MOTION 5. Forward flexion 31-60 degrees 61-90 degrees 91-120 degrees 121-150 degrees 151-180 degrees | ☐ 33<br>☐ 65<br>☐ 95<br>☐ 12 | gth of abduction (pounds) 13-15 3 |
| 7. External rotation Hand behind head, elbow Hand behind head, elbow Hand to top of head, elb Hand to top of head, elb Full elevation | w forward | nal rotation ateral thigh uttock umbosacral junction /aist (L3) 12 Vertebra terscapular (T7) |

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair

| > smith&nephe | w |
|---------------|---|
|---------------|---|


Page: 

| <pre> smith&amp;nephew <study pg="" title@master=""> xx-xxxx-xx</study></pre> | The ROWE Score for<br>Instability | Subject ID: |
|---|---|---|
| INSTRUCTIONS: Please select on | e answer from each of the following ques | stions. |
| Section 1 - Stability | | |
| ☐ No recurrence, subluxation | on or apprehension | |
| Apprehension when placi | ng arm in certain positions | |
| Subluxation (not requiring | g reduction) | |
| Recurrent dislocation | | |
| Section 2 - Motion 100% of normal ext rotation, int rotation and elevation 75% of normal ext rotation, int rotation and elevation 50% of normal ext rotation, int rotation and elevation 50% of normal elevation, and int rotation, no ext rotation | | |
| Section 3 - Function No limitation of work or sports, little or no discomfort (e.g. shoulder strong overhead, lifting, swimming, throwing, tennis Mild limitation and minimum discomfort Moderate limitation and discomfort Marked limitation and pain | | |
| With the permission of the Journal of Bone and Joint Surgery | | |

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair \*\*Smith&nephew

Number: 17-5010-06


Page: 

### 21.5 Principal Investigator Obligations (ISO 14155:2011)

#### 1. General:

a. The role of the PI is to implement and manage the day-to-day conduct of the clinical investigation as well as ensure data integrity and the rights, safety, and well-being of the subjects involved in the clinical investigation.

#### 2. Qualification of the PI. The PI shall:

- a. be qualified by education, training, and experience to assume responsibility for the proper conduct of the clinical investigation in accordance with this International Standard; evidence of such qualifications of the PI and key members of the investigation site team shall be provided to the Sponsor through up-to-date Curriculum Vitae (CV) or other relevant documentation,
- b. be experienced in the field of application and trained in the use of the investigational device under consideration,
- disclose potential conflicts of interest, including financial, that interfere with the conduct of the clinical investigation or interpretation of results, and
- d. be knowledgeable with the method of obtaining informed consent.
- 3. Qualification of investigation site. The PI shall be able to demonstrate that the proposed investigation site:
  - a. has the required number of eligible subjects needed within the agreed recruitment period, and
  - b. has one or more qualified investigators, a qualified investigation site team and adequate facilities for the foreseen duration of the clinical investigation.

#### 4. Communication with the IEC. The PI shall:

- a. provide the Sponsor with copies of any clinical-investigation-related communications between the PI and the IEC,
- b. comply with the requirements described in 4.5 of ISO 14155:2011:
  - i. Submit to the IEC the following information, any amendments and any additional documentation required by the IEC: the Protocol; IB or equivalent; informed

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




**Page:** 

consent form and any other written information provided to subjects; procedures for recruiting subjects and advertising materials, if any; a copy of the CV of the PI(s) for with the IEC has oversight.

- ii. Provide documentation of the IECs approval/favorable opinion, identifying the documents and amendments on which the opinion was based, to the Sponsor, prior to commencing the clinical investigation.
- iii. Submit the following to the IEC if required by national regulations, the protocol or IEC, whichever is more stringent:
  - 1. SAEs
  - Requests for deviations, and reports of deviations, if the deviation affects subject's rights, safety, and well-being, or the scientific integrity of the clinical investigation. Document and report to the Sponsor and IEC a report of deviations made to protect the rights, safety, and well-being of human subjects under emergency circumstances.
  - 3. Progress reports, including safety summary and deviations
  - 4. Amendments to any documents already approved by the IEC.
  - 5. If applicable, notifications of suspension or premature termination
  - 6. If applicable, justification and request for resuming the clinical investigation after suspension.
  - 7. Clinical investigation report or summary.
- iv. As a minimum, during the clinical investigation, the following information shall be obtained in writing from the IEC prior to implementation:
  - 1. Approval/favorable opinion of amendments
  - 2. Approval of the request for deviations that can affect the subject's rights, safety, and well-being or scientific integrity of the clinical investigation
  - Approval for resumption of a suspended clinical investigation if applicable.
- obtain the written and dated approval/favorable opinion of the IEC for the clinical investigation before recruiting subjects and implementing all subsequent amendments, if required,

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair




Page: 

d. promptly report any deviations from the protocol that affect the rights, safety or well-being of the subject or the scientific integrity of the clinical investigation, including those which occur under emergency circumstances, if required by the IEC, protocol or national regulations. In particular circumstances, the communication with the IEC can be performed by the Sponsor, partly or in full, in which case the Sponsor shall keep the Principal Investigator informed.

#### 5. Informed consent process. The PI shall:

#### a. General:

- Informed consent shall be obtained in writing from the subject and the process shall be documented before any procedure specific to the clinical investigation is applied to the subject; except when special circumstances for emergency treatments apply (see below)
- ii. The informed consent form consists of an information form and informed consent signature form. These two forms can either be combined in one document or separated into two documents
- b. Process of obtaining informed consent. The general process for obtaining informed consent shall be documented in the protocol and shall comply with the following. These requirements also apply with respect to informed consent obtained from a subject's legally authorized representative:
  - i. Ensure that the PI or his/her authorized designee conducts the informed consent process
  - ii. Include all aspects of the clinical investigation that are relevant to the subject's decision to participate throughout the clinical investigation
  - iii. Avoid any coercion or undue improper influence on, or inducement of, the subject to participate
  - iv. Not waive or appear to waive the subject's legal rights
  - v. Use native non-technical language that is understandable to the subject
  - vi. Provide ample time for the subject to read and understand the informed consent form and to consider participation in the clinical investigation

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06 Version: 1.0, 09/MAY/2018 Page: 

- vii. Include personally dated signatures and the PI or an authorized designee responsible for conducting the informed consent process
- viii. Show how informed consent will be obtained in special circumstances (see below) where the subject is unable to provide him or herself, and
- ix. Ensure important new information is provided to new and existing subjects throughout the clinical investigation.
- c. Special circumstances for informed consent (the following provisions are subject to national regulations):
  - i. Subject needing legally authorized representatives: informed consent may be given by the legally authorized representative only if a subject is unable to make the decision to participate in a clinical investigation (e.g. infant, child, or juvenile, seriously ill or unconscious subject, mentally ill person, mentally handicapped person). In such cases, the subject shall also be informed about the clinical investigation within his/her ability to understand.
  - ii. Subject unable to read or write: informed consent shall be obtained through a supervised oral process if a subject or legally authorized representative is unable to read or write. An independent witness shall be present throughout the process. The written informed consent form and any other information shall be read aloud and explained to the prospective subject or his/her legally authorized representative and, whenever possible, either shall sign and personally date the informed consent form. The witness also signs and personally dates the informed consent for attesting that the information was accurately explained and that the informed consent was freely given.

#### iii. Emergency treatments:

 For clinical investigations involving emergency treatments, when prior informed consent of the subject is not possible because of the subject's medical condition, the informed consent of the subject's legally authorized representative, if present, shall be requested.

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair smith&nephew


Page: 

- 2. When it is not possible to obtain prior informed consent from the subject, and the subject's legally authorized representative, is not available, the subject may still be enrolled if a specific process has been described in the protocol.
- Arrangements shall be made to inform the subject or legally authorized representative, as soon as possible, about the subject's inclusion in the clinical investigation and about all aspects of the clinical investigation.
- 4. The subject shall be asked to provide informed consent for continued participation as soon as his/her medical condition allows.
- d. The Principal Investigator may not enroll a subject without obtaining informed consent of the subject or his/her legally authorized representative only when the following conditions are fulfilled: the prospective subject fulfils the emergency conditions and is obviously in a life-threatening situation; no sufficient clinical benefits are anticipated from the currently available treatment; there is a fair possibility that the life-threatening risk to the prospective subject can be avoided if the investigational device is used; anticipated risks are outweighed by the potential benefits of applying the investigational device; the legally authorized representative cannot be promptly reached and informed.
- e. Information provided to the subject. All information pertinent to the clinical investigation, including at least the following, shall be provided in writing and in native, non-technical language that is understandable to the subject (or the subject's legally authorized representative):
  - Description and purpose
  - ii. Potential benefits
  - iii. Risks and inconveniences or the subject and, when applicable, for any embryo, foetus or nursing infant
  - iv. Alternative procedures
  - v. Confidentiality
  - vi. Compensation
  - vii. Anticipated expenses, if any, to be borne by the subject for participating in the clinical investigation

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair Number: 17-5010-06

Page: 

- viii. Information on the role of Sponsor's representative in the clinical investigation
- ix. Contact persons
- x. Statement declaring that new findings or the reasons for any amendment to the protocol that affect the subject's continued participation shall be made available to the subject.
- xi. Statement indicating that, upon the subject's approval, the subject's personal physician will be informed of the subject's participation in the clinical investigation
- xii. Termination procedures
- f. Informed consent signature shall contain the following:
  - i. The voluntary agreement to participate in the clinical investigation and follow the investigator's instructions
  - ii. A statement declaring that refusal of participation incurs no penalty for the subject
  - iii. A statement declaring that discontinuation at any time incurs no penalty for the subject
  - iv. A statement with regard to the possible consequences of withdrawal
  - v. An acknowledgement of the information provided and confirmation that all the subject's questions were answered
  - vi. A statement confirming that the subject or his/her legally authorized representative agrees to the use of the subject's relevant personal data for the purpose of the clinical investigation
  - vii. A statement confirming that the subject or his/her legally authorized representative agrees that Sponsor's representatives, regulatory authorities and IEC representatives will be granted direct access to the subject's medical records.
- g. New information: if new information becomes available that can significantly affect a subject's future health and medical care, that information shall be provided to the subject(s) affected in written form. If relevant, all affected subjects shall be asked to confirm their continuing consent in writing.
- h. ensure compliance with the applicable regulatory requirements and ethical principles for the process of obtaining informed consent, and

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



**Number:** 17-5010-06 **Version:** 1.0, 09/MAY/2018 **Page:** 

- i. ensure and document appropriate training if an authorized designee is appointed to conduct the informed consent process.
- 6. Compliance with the protocol. The Principal Investigator shall:
  - a. indicate his/her acceptance of the protocol in writing,
  - b. conduct the clinical investigation in compliance with the protocol,
  - c. create and maintain source documents throughout the clinical investigation and make them available as requested during monitoring visits or audits,
  - d. ensure that the investigational device is used solely by authorized users as specified in6.2, and in accordance with the protocol and instructions for use,
  - e. propose to the Sponsor any appropriate modification(s) of the protocol or investigational device or of the use of the investigational device,
  - f. refrain from implementing any modifications to the protocol without agreement from the Sponsor, IEC and regulatory authorities, if required,
  - document and explain any deviation from the approved protocol that occurred during the course of the clinical investigation,
  - h. ensure that an adequate investigation site team and facilities exist and are maintained and documented during the clinical investigation,
  - ensure that maintenance and calibration of the equipment relevant for the assessment of the clinical investigation is appropriately performed and documented, where applicable,
  - ensure the accuracy, completeness, legibility and timeliness of the data reported to the Sponsor in the CRF and in all required reports,
  - k. maintain the device accountability records,
  - I. allow and support the Sponsor to perform monitoring and auditing activities,
  - m. be accessible to the monitor and respond to questions during monitoring visits,
  - allow and support regulatory authorities and the IEC when performing auditing activities,
  - ensure that all clinical-investigation-related records are retained as required taking measures to prevent accidental or premature destruction, and

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair > smith&nephew


**Page:** 

- p. review and sign the clinical investigation report, as applicable.
- 7. Medical care of subjects. The Principal Investigator shall
  - a. provide adequate medical care to a subject during and after a subject's participation in a clinical investigation in the case of adverse events,
  - b. inform the subject of the nature and possible cause of any adverse events experienced,
  - c. provide the subject with the necessary instructions on proper use, handling, storage, and return of the investigational device, when it is used or operated by the subject,
  - d. inform the subject of any new significant findings occurring during the clinical investigation, including the need for additional medical care that may be required,
  - e. provide the subject with well-defined procedures for possible emergency situations
    related to the clinical investigation, and make the necessary arrangements for
    emergency treatment, including decoding procedures for blinded/masked clinical
    investigations, as needed,
  - f. ensure that clinical records are clearly marked to indicate that the subject is enrolled in a particular clinical investigation,
  - g. if appropriate, subjects enrolled in the clinical investigation shall be provided with some means of showing their participation in the clinical investigation, together with identification and compliance information for concomitant treatment measures (contact address and telephone numbers shall be provided),
  - h. inform, with the subject's approval or when required by national regulations, the subject's personal physician about the subject's participation in the clinical investigation, and
  - i. make all reasonable efforts to ascertain the reason(s) for a subject's premature withdrawal from the clinical investigation while fully respecting the subject's rights.
- 8. Safety reporting. The Principal Investigator shall:
  - a. record every adverse event and observed device deficiency, together with an assessment,

Prospective, Multicenter, Post-Market Clinical Followup Study to evaluate safety and performance of the SUTUREFIX ULTRA and SUTUREFIX CURVED Suture Anchors in shoulder and hip arthroscopic repair



Number: 17-5010-06 Version: 1.0, 09/MAY/2018 Page: 

b. report to the Sponsor, without unjustified delay, all serious adverse events and device deficiencies that could have led to a serious adverse device effect; this information shall

c) report to the IEC serious adverse events and device deficiencies that could have led
to a serious adverse device effect, if required by the national regulations or protocol or
by the IEC,

be promptly followed by detailed written reports, as specified in the protocol,

- d. report to regulatory authorities serious adverse events and device deficiencies that could have led to a serious adverse device effect, as required by the national regulations, and
- e. supply the Sponsor, upon Sponsor's request, with any additional information related to the safety reporting of a particular event.